

Certain information within this clinical study report has been redacted (ie, specific content is masked irreversibly from view with a black bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

# Statistical Analysis Plan

Study Title: A Phase 1, Open-label, Multicenter Study to Evaluate the Tolerability,

Safety, Pharmacokinetics, and Pharmacodynamics of TAK-385 Alone in Hormone Treatment-naive Japanese Patients With Non-metastatic Prostate

Cancer

Study Number: TAK-385/TB-AK160108

Sponsor: Takeda Pharmaceutical Company Limited



Version 2.0: July 20, 2017

# **Table of Contents**

| Glossary | 4 |
|---|---|
| Definition of Visit Window | 5 |
| Others | 19 |
| 1 Study Subjects, Demographics, and Other Baseline Characteristics (Part A) | 20 |
| 1.1 Disposition of Subjects | 20 |
| 1.1.1 Study Information (Part A and Part B) | 20 |
| 1.1.2 Screen Failures. | 20 |
| 1.1.3 Subject Eligibility | 21 |
| 1.1.4 Number of Subjects Who Entered the Treatment Period by Site and Treatment Group | 21 |
| 1.1.5 Disposition of Subjects | 22 |
| 1.1.6 Protocol Deviations and Analysis Sets | 23 |
| 1.2 Demographics and Other Baseline Characteristics | 24 |
| 1.2.1 Summary of Demographics and Other Baseline Characteristics | 24 |
| 1.2.2 Medical History and Concurrent Medical Conditions | 25 |
| 1.2.3 Medication History and Concomitant Medications | 25 |
| 1.3 Treatment Compliance | 26 |
| 1.3.1 Study Drug Exposure and Compliance | 26 |
| 2 Study Subjects, Demographics, and Other Baseline Characteristics (Part B) | 27 |
| 2.1 Disposition of Subjects | 27 |
| 2.1.1 Screen Failures | 27 |
| 2.1.2 Subject Eligibility | 27 |
| 2.1.3 Number of Subjects Randomized by Site and Treatment Group | 27 |
| 2.1.4 Disposition of Subjects | 28 |
| 2.1.5 Study Drug Completion Status | 29 |
| 2.1.6 Protocol Deviations and Analysis Sets | 30 |
| 2.2 Demographics and Other Baseline Characteristics | 31 |
| 2.2.1 Summary of Demographics and Other Baseline Characteristics | 31 |
| 2.2.2 Medical History and Concurrent Medical Conditions | 32 |
| 2.2.3 Medication History and Concomitant Medications | 32 |
| 2.3 Treatment Compliance | 33 |
| 2.3.1 Study Drug Exposure and Compliance | 33 |
| 2.3.2 Dosing Pattern Details | 34 |
| 3 Efficacy, Pharmacokinetic, and Pharmacodynamic Analysis (Part A) | 35 |
| 3.1 Efficacy Analysis | 35 |
| 3.1.1 Antitumor Effects | 35 |

| 3.2 Pharmacokinetic Analysis | 35 |
|---|---|
| 3.2.1 Plasma Concentrations. | 35 |
| 3.2.2 Pharmacokinetic Parameters | 35 |
| 3.3 Pharmacodynamic Analysis | 37 |
| 3.3.1 Serum Testosterone Concentrations. | 37 |
| 3.3.2 Serum Concentrations of LH, FSH, DHT, and SHBG | 37 |
| 3.4 Statistical/Analytical Issues | 37 |
| 3.4.1 Adjustments for Covariates | 37 |
| 3.4.2 Handling of Dropouts or Missing Data | 38 |
| 3.4.3 Interim Analyses and Data Monitoring | 38 |
| 3.4.4 Multicenter Studies | 38 |
| 3.4.5 Multiple Comparison/Multiplicity | 38 |
| 3.4.6 Use of an "Efficacy Subset" of Subjects | 38 |
| 3.4.7 Active-Control Studies Intended to Show Equivalence or Non-Inferiority | 38 |
| 3.4.8 Examination of Subgroups. | 38 |
| 4 Efficacy, Pharmacokinetic, and Pharmacodynamic Analysis (Part B) | 39 |
| 4.1 Efficacy Analysis | 39 |
| 4.1.1 Antitumor Effects. | 39 |
| 4.1.2 QOL Assessment | 40 |
| 4.2 Pharmacokinetic Analysis | 40 |
| 4.2.1 Plasma Concentrations. | 40 |
| 4.3 Pharmacodynamic Analysis | 41 |
| 4.3.1 Serum Testosterone Concentrations. | 41 |
| 4.3.2 Serum Concentrations of LH, FSH, DHT, and SHBG | 41 |
| 4.4 Statistical/Analytical Issues | |
| 4.4.1 Adjustments for Covariates | |
| 4.4.2 Handling of Dropouts or Missing Data | 43 |
| 4.4.3 Interim Analyses and Data Monitoring | 43 |
| 4.4.4 Multicenter Studies | 43 |
| 4.4.5 Multiple Comparison/Multiplicity | 43 |
| 4.4.6 Use of an "Efficacy Subset" of Subjects | 43 |
| 4.4.7 Active-Control Studies Intended to Show Equivalence or Non-Inferiority | 43 |
| 4.4.8 Examination of Subgroups | 43 |
| 5 Safety Analysis (Part A) | 44 |
| 5.1 Treatment-Emergent Adverse Events | 44 |
| 5.1.1 Overview of Treatment-Emergent Adverse Events | 44 |
| 5.1.2 Displays of Treatment-Emergent Adverse Events | 45 |

| 5.1.3 Displays of Dose-Limiting Toxicities | 47 |
|---|---|
| 5.2 Pretreatment Events | 47 |
| 5.2.1 Displays of Pretreatment Events | 47 |
| 5.3 Laboratory and Other Safety Data | 48 |
| 5.3.1 Laboratory Test Results | 48 |
| 5.3.2 Vital Signs, Physical Findings, and Other Observations Related to Safety | 50 |
| 5.4 Displays of Treatment-Emergent Adverse Events (Japanese) | 52 |
| 6 Safety Analysis (Part B) | 53 |
| 6.1 Treatment-Emergent Adverse Events | 53 |
| 6.1.1 Overview of Treatment-Emergent Adverse Events | 53 |
| 6.1.2 Displays of Treatment-Emergent Adverse Events | 54 |
| 6.2 Pretreatment Events | 56 |
| 6.2.1 Displays of Pretreatment Events | 56 |
| 6.3 Laboratory and Other Safety Data | 57 |
| 6.3.1 Laboratory Test Results | 57 |
| 6.3.2 Vital Signs, Physical Findings, and Other Observations Related to Safety | 60 |
| 6.4 Displays of Treatment-Emergent Adverse Events (Japanese) | 62 |
| 7 Significance Level and Confidence Coefficient (Part A and Part B) | 62 |
| Amendment History | 63 |
| Appendix 1. Amendments from the Previous Version | 1 |
| Appendix 2. Criteria for Markedly Abnormal Values and Elevated Liver Enzyme | 1 |
| Appendix 3. QOL Scoring Procedures | 1 |

#### Glossary

- Treatment-emergent adverse event (TEAE): An adverse event whose date of onset occurs on or after the start of study drug
- Descriptive statistics: number of subjects, mean, standard deviation (SD), maximum (max), minimum (min), and quartiles
- CV: coefficient of variation
- Randomized set: All subjects who were randomized. The first maintenance dose prescribed will
  be used as the treatment group when conducting analyses.
- Treatment group: For part A, the assigned cohort will be the treatment group. For part B, the first maintenance dose prescribed will be the treatment group.
- PK: pharmacokinetic
- MAV: markedly abnormal value
- ATC: anatomical therapeutic chemical
- LDH: lactic dehydrogenase
- GGT: gamma-glutamyl transpeptidase
- CK (CPK): creatine phosphokinase/kinase
- Study Day: The day before the first dose of the study drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the first dose, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.
- Follow-up Day: The day after the last dose of the study drug will be defined as Follow-up Day

  1. Follow-up Day will be calculated relative to Day 1.

#### **Definition of Visit Window**

When calculating Study Day relative to a reference date (i.e., date of first dose of study drug [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0. When calculating Study Time relative to a reference time (i.e., time of each dose of study drug), it will be calculated as: time of observation - reference time.

When calculating Follow-up Day relative to a reference date (i.e., date of last dose of study drug [Follow-up Day 0]), it will be calculated as: date of observation - reference date. Hence, reference day is always Follow-up Day 0.

All evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day/Study Time to the scheduled Study Day/Study Time will be used. If there are two observations equidistant to the scheduled Study Day/Study Time, the later observation will be used. This does not apply to the end of study visit. For the end of study visit, the last observation obtained in the corresponding time interval will be used.

<Part A>

<u>PSA</u>

| Visit | Scheduled Study Day (days) | Time Interval (days) Study Day |
|---|---|---|
| Baseline (Week 0) | Study Day: 1 | -28 - 1 |
| D28 | Study Day: 28 | 2 - 35 |

Pharmacokinetic Assessments

| Thurmdeokinette 7135e351 | | Time Interval | |
|---|---|---|---|
| Visit | Visit Scheduled Study Time (hours) | Study Day<br>(days) | Study Time<br>(hours) |
| D1 | -1 | 1 | -3.00 - 0.00 |
| D1 | 0.5 | 1 | 0.33 - 0.67 |
| D1 | 1 | 1 | 0.75 - 1.24 |
| D1 | 1.5 | 1 | 1.25 - 1.74 |
| D1 | 2 | 1 | 1.75 - 2.33 |
| D1 | 4 | 1 | 3.67 - 4.33 |
| D1 | 6 | 1 | 5.50 - 6.50 |
| D1 | 8 | 1 | 7.50 - 8.50 |
| D1 | 12 | 1 | 11.00 - 13.00 |
| D2 | -1 | 2 | -2.00 - 0.00 |
| D3 | -1 | 3 | -2.00 - 0.00 |
| D3 | 2 | 3 | 1.67 - 2.33 |
| D7 | -1 | 7 | -2.00 - 0.00 |
| D7 | 2 | 7 | 1.67 - 2.33 |
| D12 | -1 | 12 | -2.00 - 0.00 |
| D13 | -1 | 13 | -2.00 - 0.00 |
| D14 | -1 | 14 | -2.00 - 0.00 |
| D14 | 0.5 | 14 | 0.33 - 0.67 |

| | | Time Interval | |
|---|---|---|---|
| Visit | Scheduled Study Time (hours) | Study Day<br>(days) | Study Time (hours) |
| D14 | 1 | 14 | 0.75 - 1.24 |
| D14 | 1.5 | 14 | 1.25 - 1.74 |
| D14 | 2 | 14 | 1.75 - 2.33 |
| D14 | 4 | 14 | 3.67 - 4.33 |
| D14 | 6 | 14 | 5.50 - 6.50 |
| D14 | 8 | 14 | 7.50 - 8.50 |
| D14 | 12 | 14 | 11.00 - 13.00 |
| D15 | Study Day: 15 | 15 | 16.00 - 34.00<br>(from last dose) |
| D21 | Study Day: 21 | 18 - 24 | 16.00 - 34.00<br>(from last dose) |
| D28 | -1 | 28 | -2.00 - 0.00 |
| D28 | 1 | 28 | 0.75 - 1.24 |
| D28 | 2 | 28 | 1.67 - 2.33 |
| D28 | 4 | 28 | 3.67 - 4.33 |
| D28 | 8 | 28 | 7.50 - 8.50 |
| D28 | 12 | 28 | 11.00 - 13.00 |
| D29 | 24 (from D28) | 29 | 23.00 - 25.00<br>(from D28) |
| D30 | 48 (from D28) | 30 | 44.00 - 52.00<br>(from D28) |
| D31 | 72 (from D28) | 31 | 68.00 - 76.00<br>(from D28) |
| D35 | 168 (from D28) | 35 | 164.00 - 172.00<br>(from D28) |

Pharmacodynamic Assessments

| Visit | Scheduled Study Day (days) | Time Interval (days) Study Day |
|---|---|---|
| Baseline (Week 0) | Study Day: 1 | -28 - 1 |
| D2 | Study Day: 2 | 2 |
| D3 | Study Day: 3 | 3 - 4 |
| D7 | Study Day: 7 | 5 - 10 |
| D14 | Study Day: 14 | 11 - 17 |
| D21 | Study Day: 21 | 18 - 24 |
| D28 | Study Day: 28 | 25 - 29 |
| D31 | Study Day: 31 | 30 - 34 |
| D35 | Study Day: 35 | 35 |

<u>Laboratory Tests</u> (Hematology, Biochemistry, Urinalysis)

| | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | - 1 | |
| D7 | Study Day: 7 | 2 - 10 | < 15 |
| D14 | Study Day: 14 | 11 - 17 | < 15 |
| D21 | Study Day: 21 | 18 - 24 | < 15 |
| D28 | Study Day: 28 | 25 - 42 | < 15 |
| SFU | Follow-up Day: 40 | | 15 - 40 |

Laboratory Tests (Lipid and Glycated Hemoglobin in Blood)

| | Scheduled Study Day | Time Inter | val (days) |
|-------------------|---------------------|------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | - 1 | |
| D28 | Study Day: 28 | 2 - 42 | < 15 |

| | Scheduled Study Day | cheduled Study Day Time Interv | |
|-------|---------------------|--------------------------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| SFU | Follow-up Day: 40 | | 15 - 40 |

Vital Signs, Weight

| | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -28 - 1 | |
| D7 | Study Day: 7 | 2 - 10 | < 15 |
| D14 | Study Day: 14 | 11 - 17 | < 15 |
| D21 | Study Day: 21 | 18 - 24 | < 15 |
| D28 | Study Day: 28 | 25 - 42 | < 15 |
| SFU | Follow-up Day: 40 | | 15 - 40 |

12-Lead Electrocardiogram

| | Scheduled Study Day | Time Inter | val (days) |
|-------------------|---------------------|------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -28 - 1 | |
| D14 | Study Day: 14 | 2 - 20 | < 15 |
| D28 | Study Day: 28 | 21 - 42 | < 15 |
| SFU | Follow-up Day: 40 | | 15 - 40 |

**ECOG Performance Status** 

| | Scheduled Study Day<br>(days) | Time Interval (days) | |
|---|---|---|---|
| Visit | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -28 - 1 | |

# <Part B>

# **PSA**

| Visit | Scheduled Study Day (days) | Time Interval (days) Study Day |
|---|---|---|
| Baseline (Week 0) | Study Day: 1 | -28 - 1 |
| WK5D1 | Study Day: 29 | 2 - 42 |
| WK9D1 | Study Day: 57 | 43 - 70 |
| WK13D1 | Study Day: 85 | 71 - 98 |
| WK17D1 | Study Day: 113 | 99 - 126 |
| WK21D1 | Study Day: 141 | 127 - 154 |
| WK25D1 | Study Day: 169 | 155 - 210 |
| WK37D1 | Study Day: 253 | 211 - 294 |
| WK49D1 | Study Day: 337 | 295 - 378 |
| WK61D1 | Study Day: 421 | 379 - 462 |
| WK73D1 | Study Day: 505 | 463 - 546 |
| WK85D1 | Study Day: 589 | 547 - 630 |
| WK97D1 | Study Day: 673 | 631 - 680 |
| WK13D1 (LOCF) | Study Day: 85 | 2 - 98 |
| End of Study | | 2 - |

# Pharmacokinetic Assessments

| | | | Time Interval |
|---|---|---|---|
| Visit | Scheduled Study Time (hours) | Study Day<br>(days) | Study Time<br>(hours) |
| WK1D1 | -1 | 1 | -3.00 - 0.00 |
| WK1D1 | 2 | 1 | 1.75 - 2.33 |
| WK1D2 | -1 | 2 | -2.00 - 0.00 |
| WK1D4 | Study Day: 4 | 3 - 6 | 16.00 - 34.00<br>(from last dose) |

| | | Time Interval | |
|---|---|---|---|
| Visit | Visit Scheduled Study Time (hours) Study D (days) | | Study Time<br>(hours) |
| WK2D1 | Study Day: 8 | 7 - 12 | 16.00 - 34.00<br>(from last dose) |
| WK3D1 | Study Day: 15 | 13 - 22 | 16.00 - 34.00<br>(from last dose) |
| WK5D1 | Study Day: 29 | 23 - 43 | -2.00 - 0.00 |
| WK5D1 | 2 | 23 - 43 | 1.67 - 2.33 |
| WK9D1 | Study Day: 57 | 44 - 71 | 16.00 - 34.00<br>(from last dose) |
| WK13D1 | Study Day: 85 | 72 - 99 | 16.00 - 34.00<br>(from last dose) |
| WK17D1 | Study Day: 113 | 100 – 127 | 16.00 - 34.00<br>(from last dose) |
| WK21D1 | Study Day: 141 | 128 - 155 | 16.00 - 34.00<br>(from last dose) |
| WK25D1 | Study Day: 169 | 156 - 183 | 16.00 - 34.00<br>(from last dose) |
| WK37D1 | Study Day: 253 | 233 - 274 | 16.00 - 34.00<br>(from last dose) |
| WK49D1 | Study Day: 337 | 317 - 358 | 16.00 - 34.00<br>(from last dose) |

**Imaging Assessments** 

| Visit | Scheduled Study Day<br>(days) | Time Interval (days) Study Day |
|--------|-------------------------------|--------------------------------|
| WK49D1 | Study Day: 337 | 2 - 344 |
| WK97D1 | Study Day: 673 | 345 - 680 |

**QOL** Assessment

| Q O D T I SOUSSIMENT | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -28 - 1 | |
| WK5D1 | Study Day: 29 | 2 - 42 | < 15 |
| WK9D1 | Study Day: 57 | 43 - 70 | < 15 |
| WK13D1 | Study Day: 85 | 71 - 112 | < 15 |
| WK21D1 | Study Day: 141 | 113 - 154 | < 15 |
| WK25D1 | Study Day: 169 | 155 - 238 | < 15 |
| WK45D1 | Study Day: 309 | 239 - 322 | < 15 |
| WK49D1 | Study Day: 337 | 323 - 378 | < 15 |
| WK61D1 | Study Day: 421 | 379 - 462 | < 15 |
| WK73D1 | Study Day: 505 | 463 - 546 | < 15 |
| WK85D1 | Study Day: 589 | 547 - 630 | < 15 |
| WK97D1 | Study Day: 673 | 631 - 687 | < 15 |
| SFU | Follow-up Day: 40 | | 15 - 40 |

<u>Pharmacodynamic Assessments (Excluding High-Sensitivity Serum Testosterone)</u>

| Visit | Scheduled Study Day<br>(days) | Time Interval (days) Study Day |
|---|---|---|
| Baseline (Week 0) | Study Day: 1 | -28 - 1 |
| WK1D2 | Study Day: 2 | 2 - 3 |
| WK1D4 | Study Day: 4 | 4 - 5 |
| WK2D1 | Study Day: 8 | 6 - 11 |
| WK3D1 | Study Day: 15 | 12 - 21 |
| WK5D1 | Study Day: 29 | 22 - 42 |
| WK9D1 | Study Day: 57 | 43 - 70 |
| WK13D1 | Study Day: 85 | 71 - 98 |

| Visit | Scheduled Study Day<br>(days) | Time Interval (days) Study Day |
|--------|-------------------------------|--------------------------------|
| WK17D1 | Study Day: 113 | 99 - 126 |
| WK21D1 | Study Day: 141 | 127 - 154 |
| WK25D1 | Study Day: 169 | 155 - 210 |
| WK37D1 | Study Day: 253 | 211 - 294 |
| WK49D1 | Study Day: 337 | 295 - 378 |
| WK61D1 | Study Day: 421 | 379 - 462 |
| WK73D1 | Study Day: 505 | 463 - 546 |
| WK85D1 | Study Day: 589 | 547 - 630 |
| WK97D1 | Study Day: 673 | 631 - 680 |

ECOG Performance Status

| | Scheduled Study Day (days) | Time Interval (days) | |
|---|---|---|---|
| Visit | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -28 - 1 | |

Pharmacodynamic Assessments (High-Sensitivity Serum Testosterone)

| Visit | Scheduled Study Day<br>(days) | Time Interval (days) Study Day |
|---|---|---|
| Baseline (Week 0) | Study Day: 1 | -28 - 1 |
| WK2D1 | Study Day: 8 | 2 - 11 |
| WK3D1 | Study Day: 15 | 12 - 21 |
| WK5D1 | Study Day: 29 | 22 - 42 |
| WK9D1 | Study Day: 57 | 43 - 70 |
| WK13D1 | Study Day: 85 | 71 - 98 |
| WK17D1 | Study Day: 113 | 99 - 126 |
| WK21D1 | Study Day: 141 | 127 - 154 |

| Visit | Scheduled Study Day<br>(days) | Time Interval (days) Study Day |
|--------|-------------------------------|--------------------------------|
| WK25D1 | Study Day: 169 | 155 - 210 |
| WK37D1 | Study Day: 253 | 211 - 294 |
| WK49D1 | Study Day: 337 | 295 - 344 |

<u>Laboratory Tests</u> (Hematology)

| Education y Tests (Tierran | | Time Interval (days) | |
|---|---|---|---|
| Visit | Scheduled Study Day | 1 iiie iiitei | vai (uays) |
| | (days) | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | - 1 | |
| WK5D1 | Study Day: 29 | 2 - 42 | < 15 |
| WK9D1 | Study Day: 57 | 43 - 70 | < 15 |
| WK13D1 | Study Day: 85 | 71 - 126 | < 15 |
| WK25D1 | Study Day: 169 | 127 - 210 | < 15 |
| WK37D1 | Study Day: 253 | 211 - 294 | < 15 |
| WK49D1 | Study Day: 337 | 295 - 378 | < 15 |
| WK61D1 | Study Day: 421 | 379 - 462 | < 15 |
| WK73D1 | Study Day: 505 | 463 - 546 | < 15 |
| WK85D1 | Study Day: 589 | 547 - 630 | < 15 |
| WK97D1 | Study Day: 673 | 631 - 687 | < 15 |
| SFU | Follow-up Day: 40 | | 15 - 40 |

<u>Laboratory Tests (Biochemistry)</u>

| Visit | Scheduled Study Day (days) | Time Interval (days) | |
|---|---|---|---|
| | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | - 1 | |
| WK5D1 | Study Day: 29 | 2 - 42 | < 15 |
| WK9D1 | Study Day: 57 | 43 - 70 | < 15 |
| WK13D1 | Study Day: 85 | 71 - 98 | < 15 |
| WK17D1 | Study Day: 113 | 99 - 126 | < 15 |
| WK21D1 | Study Day: 141 | 127 - 154 | < 15 |
| WK25D1 | Study Day: 169 | 155 - 182 | < 15 |
| WK29D1 | Study Day: 197 | 183 - 210 | < 15 |
| WK33D1 | Study Day: 225 | 211 - 238 | < 15 |

| Visit | Scheduled Study Day (days) | Time Interval (days) | |
|--------|----------------------------|----------------------|---------------|
| | | Study Day | Follow-up Day |
| WK37D1 | Study Day: 253 | 239 - 266 | < 15 |
| WK41D1 | Study Day: 281 | 267 - 294 | < 15 |
| WK45D1 | Study Day: 309 | 295 - 322 | < 15 |
| WK49D1 | Study Day: 337 | 323 - 378 | < 15 |
| WK61D1 | Study Day: 421 | 379 - 462 | < 15 |
| WK73D1 | Study Day: 505 | 463 - 546 | < 15 |
| WK85D1 | Study Day: 589 | 547 - 630 | < 15 |
| WK97D1 | Study Day: 673 | 631 - 687 | < 15 |
| SFU | Follow-up Day: 40 | | 15 - 40 |

<u>Laboratory Tests (Lipid and Glycated Hemoglobin in Blood, Urinalysis)</u>

| Visit | Scheduled Study Day<br>(days) | Time Interval (days) | |
|---|---|---|---|
| | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | - 1 | |
| WK5D1 | Study Day: 29 | 2 - 42 | < 15 |
| WK9D1 | Study Day: 57 | 43 - 70 | < 15 |
| WK13D1 | Study Day: 85 | 71 - 126 | < 15 |
| WK25D1 | Study Day: 169 | 127 - 252 | < 15 |
| WK49D1 | Study Day: 337 | 253 - 378 | < 15 |
| WK61D1 | Study Day: 421 | 379 - 462 | < 15 |
| WK73D1 | Study Day: 505 | 463 - 546 | < 15 |
| WK85D1 | Study Day: 589 | 547 - 630 | < 15 |
| WK97D1 | Study Day: 673 | 631 - 687 | < 15 |
| SFU | Follow-up Day: 40 | | 15 - 40 |

12-Lead Electrocardiogram

| Visit | Scheduled Study Day (days) | Time Interval (days) | |
|---|---|---|---|
| | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -28 - 1 | |
| WK3D1 | Study Day: 15 | 2 - 21 | < 15 |
| WK5D1 | Study Day: 29 | 22 - 98 | < 15 |
| WK25D1 | Study Day: 169 | 99 – 252 | < 15 |
| WK49D1 | Study Day: 337 | 253 – 420 | < 15 |
| WK73D1 | Study Day: 505 | 421 – 588 | < 15 |
| WK97D1 | Study Day: 673 | 589 - 687 | < 15 |
| SFU | Follow-up Day: 40 | | 15 - 40 |

Vital Signs, Weight

| Visit | Scheduled Study Day<br>(days) | Time Interval (days) | |
|---|---|---|---|
| | | Study Day | Follow-up Day |
| Baseline (Week 0) | Study Day: 1 | -28 - 1 | |
| WK2D1 | Study Day: 8 | 2 - 11 | < 15 |
| WK3D1 | Study Day: 15 | 12 - 21 | < 15 |
| WK5D1 | Study Day: 29 | 22 - 42 | < 15 |
| WK9D1 | Study Day: 57 | 43 - 70 | < 15 |
| WK13D1 | Study Day: 85 | 71 - 126 | < 15 |
| WK25D1 | Study Day: 169 | 127 - 252 | < 15 |
| WK49D1 | Study Day: 337 | 253 - 378 | < 15 |
| WK61D1 | Study Day: 421 | 379 - 462 | < 15 |
| WK73D1 | Study Day: 505 | 463 - 546 | < 15 |
| WK85D1 | Study Day: 589 | 547 - 630 | < 15 |
| WK97D1 | Study Day: 673 | 631 - 687 | < 15 |
| SFU | Follow-up Day: 40 | | 15 - 40 |

# Bone Mineral Density (DXA)

| Visit | Scheduled Study Day (days) | Time Interval (days) Study Day |
|---|---|---|
| Baseline (Week 0) | Study Day: 1 | -28 - 1 |
| WK25D1 | Study Day: 169 | 2 - 252 |
| WK49D1 | Study Day: 337 | 253 - 420 |
| WK73D1 | Study Day: 505 | 421 - 588 |
| WK97D1 | Study Day: 673 | 589 - 713 |

#### **Others**

- Duration of exposure to study drug (days): date of last dose of study drug date of first dose of study drug + 1
- Dose intensity (mg/day): total amount of doses taken / duration of exposure to study drug (rounded to 1 decimal place)
- Relative dose intensity (%): (total amount of doses taken / total dose expected per initial dose) \*
   100 (rounded to 1 decimal place)
- Dosing compliance: (total amount of doses taken / total dose expected) \* 100 (rounded to 1 decimal place)
- Disease duration (days): date subject signed Informed Consent Form date of diagnosis + 1
  - For the date subject signed Informed Consent Form, the year, the month, and the day will be used for the calculation.
  - ➤ If the year is unknown, then the date of diagnosis will be treated as missing. If the month is unknown, then the month will be treated as January and the day will be treated as the 1<sup>st</sup> day of the month. If only the day is unknown, then the day will be treated as the 1<sup>st</sup> day of the month for the calculation.

#### • PK parameters:

- ➤ AUC<sub>last</sub> --Area under the concentration-time curve from time 0 to time of the last quantifiable concentration.
- ➤ AUC<sub>last, ss</sub> --Area under the concentration-time curve from time 0 to time of the last quantifiable concentration, at steady state.
- $\triangleright$  AUC<sub> $\tau$ </sub> --Area under the concentration-time curve during a dosing interval (= 24 hours).
- ightharpoonup AUC<sub> $\tau$ , ss</sub> --Area under the concentration-time curve during a dosing interval (= 24 hours), at steady state.
- ightharpoonup AUC<sub> $\tau$ , ss</sub>/D --Dose-normalized AUC<sub> $\tau$ </sub>, at steady state.
- CL/F<sub>ss</sub> --Apparent clearance after extravascular administration, at steady state, calculated using AUC<sub>τ</sub>.
- ➤ C<sub>max</sub> --Maximum observed concentration.
- C<sub>max, ss</sub> --Maximum observed concentration, at steady state.
- $ightharpoonup C_{max, ss}/D$  --Dose-normalized  $C_{max}$ , at steady state.
- > C<sub>min, ss</sub> --Minimum observed concentration during a dosing interval, at steady state.
- $\lambda_z$  --Terminal disposition phase rate constant.
- ightharpoonup t<sub>max</sub> --Time of first occurrence of C<sub>max</sub>.
- $\succ$  t<sub>max, ss</sub> --Time of first occurrence of C<sub>max</sub>, at steady state.
- ightharpoonup t<sub>1/2z</sub> --Terminal disposition phase half-life.
- V<sub>z</sub>/F<sub>ss</sub> --Apparent volume of distribution during the terminal disposition phase after extravascular administration, calculated using AUC<sub>τ</sub>.

## 1 Study Subjects, Demographics, and Other Baseline Characteristics (Part A)

### 1.1 Disposition of Subjects

## 1.1.1 Study Information (Part A and Part B)

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version
WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical

Method(s): (1) Study Information

Study information shown in the analysis variables section will be provided.

#### 1.1.2 Screen Failures

Analysis Set: All Subjects Who Did Not Enter the Treatment Period

Analysis

Variable(s): Age (years) [Min<= - <= 64, 65<= - <= 74,

 $75 \le - \le Max$ 

Gender [Male, Female]

Analytical

Method(s): (1) Screen Failures

Frequency distributions for categorical variables and descriptive statistics for

continuous variables will be provided.

## 1.1.3 Subject Eligibility

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis Eligibility Status [Eligible for Entrance into the

Variable(s): Treatment Period, Not Eligible for

Entrance into the Treatment Period

Primary Reason for Subject Not [Pretreatment Event/Adverse Event,

Being Eligible Major Protocol Deviation, Lost to

Follow-Up, Voluntary Withdrawal, Study Termination, Did Not Meet

Entrance Criteria, Other]

Analytical

Method(s): (1) Eligibility for Entrance into the Treatment Period

Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being eligible, the total number of

ineligible subjects will be used as the denominator.

1.1.4 Number of Subjects Who Entered the Treatment Period by Site and Treatment Group

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

Variable(s): Status of Entrance into the [Entered]

**Treatment Period** 

Stratum: Site [Site numbers will be used as categories]

Analytical

Method(s): (1) Number of Subjects Who Entered the Treatment Period by Site and

Treatment Group

Frequency distribution will be provided for each stratum by treatment group

and overall.

#### 1.1.5 Disposition of Subjects

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

Variable(s): Study Drug Administration Status [Eligible but Not Treated]

Reason for Not Being Treated [Pretreatment Event/Adverse Event,

Major Protocol Deviation, Lost to Follow-Up, Voluntary Withdrawal, Study Termination, Lack of Efficacy,

Other]

Study Drug Completion Status [Completed Study Drug, Prematurely

Discontinued Study Drug]

Reason for Discontinuation of

Study Drug

[Pretreatment Event/Adverse Event,

Major Protocol Deviation, Lost to Follow-Up, Voluntary Withdrawal,

Study Termination, Lack of Efficacy,

Other]

Completion Status of the Safety

Follow-up

[Completed Safety Follow-up,

Prematurely Discontinued Safety

Follow-up]

Reason for Discontinuation of the

Safety Follow-up

[Pretreatment Event/Adverse Event,

Major Protocol Deviation, Lost to

Follow-Up, Voluntary Withdrawal,

Study Termination, Lack of Efficacy,

Other]

Analytical

Method(s):

(1) Disposition of Subjects

Frequency distributions will be provided for each treatment group and overall. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation of study drug, the total number of subjects who prematurely discontinued the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation of the safety follow-up, the total number of subjects who prematurely discontinued the safety follow-up will be used as the denominator.

#### 1.1.6 Protocol Deviations and Analysis Sets

#### 1.1.6.1 Protocol Deviations

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

Variable(s): Protocol Deviation [Major GCP Violations, Deviations of Protocol

Entry Criteria, Deviations of Discontinuation Criteria, Deviations Related to Treatment Procedure or Dose, Deviations Concerning Excluded Medication or Therapy, Deviations to

Avoid Emergency Risk]

Analytical

Method(s): (1) Protocol Deviations

Frequency distribution will be provided by treatment group and overall for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

#### 1.1.6.2 Analysis Sets

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

Variable(s): Handling of Subjects and Subject Data [Categories are based on the

specifications in Handling

Rules for Analysis Data]

**Analysis Sets** 

Full Analysis Set [Included]
Safety Analysis Set [Included]
DLT Analysis Set [Included]
Pharmacokinetic Analysis Set [Included]

Analytical

Method(s): (1) Subjects Excluded from Analysis Sets

(2) Subject Data Excluded from Analysis Sets

(3) Analysis Sets

Frequency distributions will be provided by treatment group for (1) and (2) and by treatment group and overall for (3). For (1) and (2), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

#### 1.2 Demographics and Other Baseline Characteristics

## 1.2.1 Summary of Demographics and Other Baseline Characteristics

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Age (years) [Min<= - <=64, 65<= - <=74,

 $75 \le - \le Max$ 

Gender [Male, Female]

Height (cm)

Weight (kg) (Week 0) BMI (kg/m<sup>2</sup>) (Week 0)

Smoking Classification [The subject has never smoked,

The subject is a current smoker,

The subject is an ex-smoker]

ECOG Performance Status (Week

[0, 1, 2, 3, 4]

0)

Diagnostic Method [Histological Diagnosis, Cytological

Diagnosis, Other]

Disease Duration (days)

Gleason Grading System (Gleason [2, 3, 4, 5, 6

[2, 3, 4, 5, 6, 7, 8, 9, 10]

Score)

Histologic Type [Adenocarcinoma, Other]

Degree of Differentiation [Well Differentiated

Adenocarcinoma, Moderately

Differentiated Adenocarcinoma,

Poorly Differentiated Adenocarcinoma,

Unclassified Adenocarcinoma]

TNM Classification T [T0, T1, T2, T3, T4, TX]

TNM Classification N [N0, N1, NX]
TNM Classification M [M0, M1, MX]

Prostatectomy [Yes, No]

Radical Prostatectomy [Yes, No]

High-Intensity Focused Ultrasound [Yes, No]
Radiation Therapy [Yes, No]
Other Treatment [Yes, No]

PSA (ng/mL) (Week 0)

Testosterone (ng/mL) (Week 0)

Analytical

Method(s): (1) Summary of Demographics and Baseline Characteristics

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided by treatment group and overall.

## 1.2.2 Medical History and Concurrent Medical Conditions

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Medical History

**Concurrent Medical Conditions** 

Analytical

Method(s): (1) Medical History by System Organ Class and Preferred Term

(2) Concurrent Medical Conditions by System Organ Class and Preferred

Term

Frequency distributions will be provided for each treatment group and overall. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

#### 1.2.3 Medication History and Concomitant Medications

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Medication History

**Concomitant Medications** 

Analytical

Method(s): (1) Medication History by Preferred Medication Name

(2) Concomitant Medications That Started Prior to and Were Ongoing at Baseline as well as Those That Started After Baseline by ATC

Pharmacological Subgroup and Preferred Medication Name

Frequency distributions will be provided for each treatment group and overall. WHO Drug dictionary will be used for coding. Summaries will be provided using preferred medication names for (1) and using both ATC pharmacological subgroup and preferred medication names for (2). ATC

pharmacological subgroup will be sorted alphabetically and preferred medication names will be sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication name will be counted only once for that preferred medication name.

### 1.3 Treatment Compliance

## 1.3.1 Study Drug Exposure and Compliance

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Duration of Exposure to Study Drug [1<= - <= 7, 8<= - <= 14, 15<= - <= 21,

(days) 22 <= - <= Max]

Total Amount of Doses Taken (mg)

Dose Intensity (mg/day) Relative Dose Intensity (%)

Subjects with Any Dose Held [Yes, No]

Reason for Dose Being Held

Adverse Event [Yes]

Other [Yes]

Dosing Compliance (%) [Min<= - <=79.9, 80.0<= - <=89.9,

 $90.0 \le - \le Max$ 

Analytical

Method(s): (1) Study Drug Exposure and Compliance

Frequency distributions for categorical variables and descriptive statistics for

continuous variables will be provided by treatment group and overall.

### 2 Study Subjects, Demographics, and Other Baseline Characteristics (Part B)

## 2.1 Disposition of Subjects

#### 2.1.1 Screen Failures

Analysis Set: All Subjects Who Were Not Randomized

Analysis

Variable(s): Age (years) [Min<= - <=64, 65<= - <=74,

 $75 \le - \le Max$ 

Gender [Male, Female]

Analytical

Method(s): (1) Screen Failures

Frequency distributions for categorical variables and descriptive statistics for

continuous variables will be provided.

2.1.2 Subject Eligibility

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis Eligibility Status [Eligible for Randomization, Not Eligible for

Variable(s): Randomization]

Primary Reason for [Pretreatment Event/Adverse Event, Major Subject Not Being Eligible Protocol Deviation, Lost to Follow-Up,

Voluntary Withdrawal, Study Termination,

Did Not Meet Entrance Criteria, Other]

Analytical

Method(s): (1) Eligibility for Randomization

Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being eligible, the total number of

ineligible subjects will be used as the denominator.

2.1.3 Number of Subjects Randomized by Site and Treatment Group

Analysis Set: Randomized Set

Analysis

Variable(s): Randomization Status [Randomized]

Stratum: Site [Site numbers will be used as categories]

Analytical

Method(s): (1) Number of Subjects Randomized by Site and Treatment Group

Frequency distribution will be provided for each stratum by treatment group

and overall.

## 2.1.4 Disposition of Subjects

Analysis Set: Randomized Set

Subjects from the Randomized Set Who Completed Study Drug (48 Weeks)

Analysis

Variable(s): Study Drug Administration Status [Randomized but Not Treated]

Reason for Not Being Treated [Pretreatment Event/Adverse Event,

Major Protocol Deviation, Lost to Follow-Up, Voluntary Withdrawal, Study Termination, Lack of Efficacy,

Other]

Study Drug Completion Status (48

Weeks)

[Completed Study Drug (48 Weeks),

Prematurely Discontinued Study

Drug (48 Weeks)]

Reason for Discontinuation of

Study Drug

[Pretreatment Event/Adverse Event, Major Protocol Deviation, Lost to Follow-Up, Voluntary Withdrawal, Study Termination, Lack of Efficacy,

Other]

Entrance into the Extension

**Treatment Period** 

[Entered the Extension Treatment

Period, Did Not Enter the Extension

Treatment Period]

Reason for Not Entering the

**Extension Treatment Period** 

[Pretreatment Event/Adverse Event,

Major Protocol Deviation, Lost to

Follow-Up, Voluntary Withdrawal, Study Termination, Lack of Efficacy,

Start of Other Treatment, Other]

Study Drug Completion Status (96

Weeks)

[Completed Study Drug (96 Weeks),

Prematurely Discontinued Study

Drug (96 Weeks)]

Reason for Discontinuation of

Study Drug

[Pretreatment Event/Adverse Event,

Major Protocol Deviation, Lost to Follow-Up, Voluntary Withdrawal,

Study Termination, Lack of Efficacy,

Completed 48 Weeks of Treatment but Did Not Enter Extension, Other]

Completion Status of the Safety [Completed Safety Follow-up,

Follow-up Prematurely Discontinued Safety

Follow-up]

Reason for Discontinuation of the [Pr

Safety Follow-up

[Pretreatment Event/Adverse Event, Major Protocol Deviation, Lost to

Follow-Up, Voluntary Withdrawal,

Study Termination, Lack of Efficacy,

Other]

Analytical

Method(s): (1) Disposition of Subjects

Randomized set will be used to perform the following analysis, with the exception of the summary for entrance into the extension treatment period and the reasons for not entering which will use subjects from the randomized set who completed study drug (48 weeks). Frequency distributions will be provided for each treatment group and overall. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation at 48 weeks and 96 weeks, the total number of subjects who prematurely discontinued the study drug before 48 weeks and 96 weeks (including subjects who completed 48 weeks of study drug treatment but did not enter the extension treatment period), respectively, will be used as the denominator. When calculating percentages for the reasons for not entering the extension treatment period, the total number of subjects who completed 48 weeks of study drug treatment but did not enter the extension treatment period will be used as the denominator.

### 2.1.5 Study Drug Completion Status

Analysis Set: Randomized Set

Analysis Study Drug Completion Status (96 [Completed Study Drug (96 Weeks),

Variable(s): Weeks) Prematurely Discontinued Study

Drug (96 Weeks)]

Reason for Discontinuation of

Study Drug

[Pretreatment Event/Adverse Event, Major Protocol Deviation, Lost to Follow-Up, Voluntary Withdrawal, Study Termination, Lack of Efficacy, Completed 48 Weeks of Treatment but Did Not Enter Extension, Other] Categories: Duration of Exposure to Study Drug  $[0 \le - \le 90, 91 \le - \le 180,$ 

(days) 181<= - <=270, 271<= - <=360,

361<= - <=450, 451<= - <=540,

 $541 \le - \le 630, 631 \le - \le Max$ 

Analytical

Method(s): (1) Study Drug Completion Status

Frequency distribution will be provided for each category of duration of

exposure to study drug by treatment group and overall.

## 2.1.6 Protocol Deviations and Analysis Sets

#### 2.1.6.1 Protocol Deviations

Analysis Set: Randomized Set

Analysis

Variable(s): Protocol Deviation [Major GCP Violations, Deviations of Protocol

Entry Criteria, Deviations of Discontinuation Criteria, Deviations Related to Treatment Procedure or Dose, Deviations Concerning

Excluded Medication or Therapy, Deviations to

Avoid Emergency Risk]

Analytical

Method(s): (1) Protocol Deviations

Frequency distribution will be provided by treatment group and overall for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that

can be classified into the same category will be counted only once.

### 2.1.6.2 Analysis Sets

Analysis Randomized Set

Set:

Analysis

Variable(s): Handling of Subjects and Subject Data [Categories are based on the

specifications in Handling Rules for

Analysis Data]

Analysis Sets

Full Analysis Set [Included]
Safety Analysis Set [Included]
Pharmacokinetic Analysis Set [Included]

Analytical

Method(s): (1) Subjects Excluded from Analysis Sets

(2) Subject Data Excluded from Analysis Sets

(3) Analysis Sets

Frequency distributions will be provided by treatment group for (1) and (2) and by treatment group and overall for (3). For (1) and (2), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

## 2.2 Demographics and Other Baseline Characteristics

# 2.2.1 Summary of Demographics and Other Baseline Characteristics

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Age (years) [Min<= - <= 64, 65<= - <= 74,

 $75 \le - \le Max$ 

Gender [Male, Female]

Height (cm)

Weight (kg) (Week 0) BMI (kg/m<sup>2</sup>) (Week 0)

Smoking Classification [The subject has never smoked,

The subject is a current smoker,

The subject is an ex-smoker]

ECOG Performance Status (Week 0) [0, 1, 2, 3, 4]

Diagnostic Method [Histological Diagnosis, Cytological

Diagnosis, Other]

Disease Duration (days)

Gleason Grading System (Gleason [2, 3, 4, 5, 6, 7, 8, 9, 10]

Score)

Histologic Type [Adenocarcinoma, Other]

Degree of Differentiation [Well Differentiated

Adenocarcinoma, Moderately

Differentiated Adenocarcinoma,

Poorly Differentiated

Adenocarcinoma, Unclassified

Adenocarcinoma]

TNM Classification T [T0, T1, T2, T3, T4, TX]

TNM Classification N [N0, N1, NX]

TNM Classification M [M0, M1, MX]

Prostatectomy [Yes, No]

Radical Prostatectomy [Yes, No]

High-Intensity Focused Ultrasound [Yes, No]

Radiation Therapy [Yes, No]

Other Treatment [Yes, No]

PSA (ng/mL) (Week 0)

Testosterone (ng/mL) (Week 0)

Analytical

Method(s): (1) Summary of Demographics and Baseline Characteristics

Frequency distributions for categorical variables and descriptive statistics for

continuous variables will be provided by treatment group and overall.

### 2.2.2 Medical History and Concurrent Medical Conditions

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Medical History

**Concurrent Medical Conditions** 

Analytical

Method(s): (1) Medical History by System Organ Class and Preferred Term

(2) Concurrent Medical Conditions by System Organ Class and Preferred

Term

Frequency distributions will be provided for each treatment group and overall. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

## 2.2.3 Medication History and Concomitant Medications

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Medication History

**Concomitant Medications** 

Analytical

Method(s): (1) Medication History by Preferred Medication Name

(2) Concomitant Medications That Started Prior to and Were Ongoing at
Baseline as well as Those That Started After Baseline by ATC
Pharmacological Subgroup and Preferred Medication Name
Frequency distributions will be provided for each treatment group and
overall. WHO Drug dictionary will be used for coding. Summaries will be
provided using preferred medication names for (1) and using both ATC
pharmacological subgroup and preferred medication names for (2). ATC
pharmacological subgroup will be sorted alphabetically and preferred
medication names will be sorted in decreasing frequency based on the
number of reports. A subject who has been administered several medications
with the same preferred medication name will be counted only once for that
preferred medication name.

### 2.3 Treatment Compliance

# 2.3.1 Study Drug Exposure and Compliance

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Duration of Exposure to Study Drug [1<= - <=90, 91<= - <=180,

(days) 181<= - <=270, 271<= - <=360,

361<= - <=450, 451<= - <=540,

541<= - <=630, 631<= - <=Max]

Total Amount of Doses Taken (mg)

Dose Intensity (mg/day)

Relative Dose Intensity (%)

Subjects with Any Dose Held [Yes, No]

Reason for Dose Being Held

Adverse Event [Yes]

Other [Yes]

Subjects with Any Dose Reduction [Yes, No]

Reason for Dose Being Reduced

Adverse Event [Yes]

Other [Yes]

Dosing Compliance (%) [Min<= - <=79.9, 80.0<= - <=89.9,

 $90.0 \le - \le Max$ 

Analytical

Method(s): (1) Study Drug Exposure and Compliance

Frequency distributions for categorical variables and descriptive statistics for

continuous variables will be provided by treatment group and overall.

# 2.3.2 Dosing Pattern Details

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Dosing Pattern [80 mg,

120 mg,

80 / 120 mg,

80 / 120 / 80 mg,

80 / 40 mg,

120 / 160 mg,

120 / 160 / 120 mg,

120 / 80 mg, etc.]

\*These categories are merely an

example and may change in

accordance with the actual data.

Last Dose [40 mg, 80 mg, 120 mg, 160 mg]

Analytical

Method(s): (1) Dosing Pattern Details

Frequency distributions will be provided by treatment group and overall.
## 3 Efficacy, Pharmacokinetic, and Pharmacodynamic Analysis (Part A)

## 3.1 Efficacy Analysis

#### 3.1.1 Antitumor Effects

Analysis Set: Full Analysis Set

Analysis

Variable(s): PSA (ng/mL)
Visit: Baseline, D28

Analytical

Method(s): The following analysis will be performed using the full analysis set.

For the observed values, descriptive statistics and two-sided 95% confidence intervals of the mean will be provided for each visit by treatment group. The same analysis will be performed for the percent change from baseline.

### 3.2 Pharmacokinetic Analysis

### 3.2.1 Plasma Concentrations

Analysis Set: Pharmacokinetic Analysis Set

Analysis

Variable(s): Plasma concentrations of TAK-385 (ng/mL)

Visit: D1 and D14: Before dosing, 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours after dosing

D28: Before dosing, 1, 2, 4, 8, 12, 24, 48 and 72 hours after dosing

D3 and D7: Before dosing and 2 hours after dosing D2, D12, D13, D15, D21 and D35: Before dosing

Analytical Number of subjects, mean, SD, min, median, max, geometric mean, and CV

Method(s): will be used to summarize plasma concentrations at each visit for each

treatment group.

Linear plots of plasma concentration-time profiles will be provided for each treatment group using individual and mean (SD) concentrations in separate plots. Mean (SD) plots will include the plasma concentration plot for all visits, separate plots for each of Day 1, Day 14, Day 28, and a plot for the

plasma trough concentrations.

#### 3.2.2 Pharmacokinetic Parameters

Listing

Analysis Set: Full Analysis Set

Analysis

Variable(s): D1:  $AUC_{\tau}$ ,  $C_{max}$  and  $t_{max}$ 

D14:  $AUC_{last, ss}$ ,  $AUC_{\tau, ss}$ ,  $AUC_{\tau, ss}$ /D,  $C_{max, ss}$ ,  $C_{max, ss}$ /D,  $C_{min, ss}$ ,  $t_{max, ss}$ 

D28:  $AUC_{last, ss}$ ,  $AUC_{\tau, ss}$ ,  $AUC_{\tau, ss}$ /D,  $CL/F_{ss}$ ,  $C_{max, ss}$ ,  $C_{max, ss}$ /D,  $t_{max, ss}$ ,  $t_{1/2z}$ ,  $V_z/F_{ss}$ ,  $\lambda_z$ , number of data points with first and last data points used in the terminal disposition phase regression analysis and adjusted  $R^2$  (coefficient of determination) for the terminal disposition phase regression analysis

Analytical

Method(s):

PK parameters will be calculated by using individual plasma concentrations with actual sampling times. Plasma concentrations from D1 to D2, D14 to D15 and D28 to D35 will be used for the calculation of PK parameters on D1, D14 and D28 respectively. Plasma concentrations deviated from the visit window will be also used for the calculation. A standard non-compartmental analysis will be performed using the linear trapezoidal rule. If subject received prohibited concomitant medications, therapies or foods, then the plasma concentrations measured on and after this day will be used to estimate the PK parameters for the listing but the results will be treated as reference values.

Individual PK parameters will be listed. The listings will include the treatment group, subject ID and evaluation day (D1, D14, and D28) in addition to the PK parameters.

#### **Descriptive Statistics**

Analysis Set: Pharmacokinetic Analysis Set

Analysis D1:  $AUC_{\tau}$ ,  $C_{max}$  and  $t_{max}$ 

 $Variable(s): \quad D14: \quad AUC_{last, \, ss}, \, AUC_{\tau, \, ss}, \, AUC_{\tau, \, ss}/D, \, C_{max, \, ss}, \, C_{max, \, ss}/D, \, C_{min, \, ss}, \, t_{max, \, ss}$ 

 $D28: \quad AUC_{last, \, ss}, \, AUC_{\tau, \, ss}, \, AUC_{\tau, \, ss}/D, \, CL/F_{ss}, \, C_{max, \, ss}, \, C_{max, \, ss}/D, \, t_{max, \, ss} \; , \, t_{1/2z}, \, t_{max, \, ss} \; , \,$ 

 $V_z/F_{ss}$ ,  $\lambda_z$ 

Analytical

Method(s):

For the pharmacokinetic parameters, the number of subjects, mean, SD, min, median, max, geometric mean, and CV will be provided for each treatment group. PK parameters which are treated as reference values will be excluded from the summary statistics.

Graphical assessment of dose-proportionality on  $C_{max, ss}$  and  $AUC_{\tau, ss}$  will be conducted on D14 and D28 by plotting individual dose-normalized exposure parameters, i.e.,  $C_{max, ss}/D$  or  $AUC_{\tau, ss}/D$  versus dose.

### 3.3 Pharmacodynamic Analysis

#### 3.3.1 Serum Testosterone Concentrations

Analysis Set: Full Analysis Set

Analysis

Variable(s): Serum Testosterone Concentrations (ng/mL)

Visit: Baseline, D2, D3, D7, D14, D21, D28, D31, D35

Analytical

Method(s): The following analysis will be performed using the full analysis set.

For observed values and percent change from baseline, descriptive statistics and two-sided 95% confidence intervals of the mean will be provided for each visit by treatment group. Case plots as well as the mean and standard deviation plots of changes over time will be provided for observed values for each treatment group. A reference line will be drawn where the serum

testosterone concentration is 0.5 ng/mL.

### 3.3.2 Serum Concentrations of LH, FSH, DHT, and SHBG

Analysis Set: Full Analysis Set

Analysis

Variable(s): (1) Serum Concentrations of LH (mIU/mL)

(2) Serum Concentrations of FSH (mIU/mL)

(3) Serum Concentrations of DHT (ng/mL)

(4) Serum Concentrations of SHBG (nmol/L)

Visit: Baseline, D2, D3, D7, D14, D21, D28, D31, D35

Analytical

Method(s): The following analysis will be performed using the full analysis set.

For the analysis variables (1) to (4), descriptive statistics of the observed values and the two-sided 95% confidence intervals of the mean will be provided for each visit by treatment group. The same analysis will be performed for the percent change from baseline. Case plots as well as the mean and standard deviation plots of changes over time will be provided for

observed values for each treatment group.

## 3.4 Statistical/Analytical Issues

#### 3.4.1 Adjustments for Covariates

Not applicable in this study.

### 3.4.2 Handling of Dropouts or Missing Data

Missing test results and data determined to be non-evaluable according to the Handling Rules for Analysis Data will not be used for hypothesis testing and estimations.

Values less than or equal to the lower limit of quantification will be treated as the value of the lower limit of quantification for PSA, serum testosterone, LH, FSH, DHT, and SHBG, and all others will be treated as zero when calculating the descriptive statistics.

Values less than the lower limit of quantification will be treated as zero except for the calculation of geometric mean for plasma concentration of TAK-385. For the geometric mean, values less than the lower limit of quantification will be treated as missing.

## 3.4.3 Interim Analyses and Data Monitoring

No interim analysis is planned in this study.

#### 3.4.4 Multicenter Studies

Although this study is a multicenter study, treatment-by-center interaction will not be explored since the number of subjects for each center is not sufficient for such exploration.

## 3.4.5 Multiple Comparison/Multiplicity

Not applicable in this study.

## 3.4.6 Use of an "Efficacy Subset" of Subjects

Not applicable in this study.

## 3.4.7 Active-Control Studies Intended to Show Equivalence or Non-Inferiority

Not applicable in this study.

## 3.4.8 Examination of Subgroups

Not applicable in this study.

#### 4 Efficacy, Pharmacokinetic, and Pharmacodynamic Analysis (Part B)

## 4.1 Efficacy Analysis

### 4.1.1 Antitumor Effects

Analysis Set: Full Analysis Set

Analysis

Variable(s): (1) PSA (ng/mL)

(2) Rate of Progression Based on PSA (%)

(3) Rate of Progression Based on Imaging Assessments (%)

Visit: (1) Baseline, WK5D1, WK9D1, WK13D1, WK17D1, WK21D1, WK25D1,

WK37D1, WK49D1, WK61D1, WK73D1, WK85D1, WK97D1,

WK13D1 (LOCF), End of Study

(3) WK49D1, WK97D1

Analytical

Method(s): The following analysis will be performed using the full analysis set.

(1) For the observed values, descriptive statistics and two-sided 95% confidence intervals of the mean will be provided for each visit by treatment group. Case plots as well as the mean and standard deviation plots of changes over time will be provided for each treatment group. The same analysis will be performed for the percent change from baseline.

The percent change from baseline at WK13D1 (LOCF) as well as the percent change from baseline when the PSA value is at its minimum since the start of the study drug administration will be shown using waterfall plots for each treatment group.

- (2) Rate of progression based on PSA will be defined as the proportion of subjects who have a 25% or greater increase as well as an absolute increase of 2 ng/mL or more in the value of PSA at least 4 weeks from the nadir. If the value of PSA never decreased from baseline, the above conditions will be fit to the value obtained after WK13D1. A missing value will be assigned if neither of the following conditions is met: "there are at least two observations after study drug administration" or "there is at least one observation on or after WK13D1 and the baseline is not missing". If the same minimum PSA value occurs at several visits, then the PSA value with the earliest date will be used as the nadir. Frequency distributions will be provided for each treatment group.
- (3) Rate of progression based on imaging assessments will be defined as the proportion of subjects who have developed new lesions. Frequency distributions will be provided for each visit by treatment group.

#### 4.1.2 OOL Assessment

Analysis Set: Full Analysis Set

Analysis

Variable(s): (1) AMS

(2) EORTC-QLQ-C30

(3) EPIC

Visit: Baseline, WK5D1, WK9D1, WK13D1, WK21D1, WK25D1, WK45D1,

WK49D1, WK61D1, WK73D1, WK85D1, WK97D1, SFU

Analytical

 $Method(s): \qquad \text{The following analysis will be performed using the full analysis set. The} \\$ 

scoring procedures are described in detail in the Appendix.

(1) Descriptive statistics for the actual values and the percent change from baseline of AMS subscale scores and total scores will be provided for each

visit by treatment group.

(2) Descriptive statistics for the actual values and the change from baseline of

Global health status/QoL score and each Functional scales score (physical,

role, emotional, cognitive, social) will be provided for each visit by treatment

group.

(3) Descriptive statistics for the actual values and the change from baseline of

each HRQOL Domain Summary Score (urinary, bowel, sexual, hormonal)

will be provided for each visit by treatment group.

#### 4.2 Pharmacokinetic Analysis

#### **4.2.1 Plasma Concentrations**

Analysis Set: Pharmacokinetic Analysis Set

Analysis

Variable(s): Plasma concentrations of TAK-385 (ng/mL)

Visit: WK1D1 and WK5D1: Before dosing and 2 hours after dosing.

WK1D2, WK1D4, WK2D1, WK3D1, WK9D1, WK13D1, WK17D1,

WK21D1, WK25D1, WK37D1 and WK49D1: Before dosing

Analytical

Method(s): Descriptive statistics, geometric mean, and CV will be used to summarize

plasma concentrations at each visit for each treatment group.

Case plots as well as the mean and standard deviation plots of changes over

time will be provided for plasma concentrations for each treatment group.

### 4.3 Pharmacodynamic Analysis

#### 4.3.1 Serum Testosterone Concentrations

Analysis Set: Full Analysis Set

Analysis

Variable(s): (1) Serum Testosterone Concentrations (ng/mL)

(2) High-sensitivity Serum Testosterone Concentrations (ng/dL)

(3) Castration Rate (%)

Visit: (1) Baseline, WK1D2, WK1D4, WK2D1, WK3D1, WK5D1, WK9D1,

WK13D1, WK17D1, WK21D1, WK25D1, WK37D1, WK49D1,

WK61D1, WK73D1, WK85D1, WK97D1

(2) Baseline, WK2D1, WK3D1, WK5D1, WK9D1, WK13D1, WK17D1,

WK21D1, WK25D1, WK37D1, WK49D1

Analytical

Method(s): The following analysis will be performed using the full analysis set.

For the analysis variables (1) and (2), descriptive statistics and two-sided 95% confidence intervals of the mean will be provided for the observed values and the percent change from baseline for each visit by treatment

group. Case plots as well as the mean and standard deviation plots of changes

over time will be provided for observed values for each treatment group. For

(1), a reference line will be drawn where the serum testosterone concentration

is 0.5 ng/mL.

(3) Castration rate will be defined as the proportion of subjects who have

serum testosterone concentrations of less than 0.5 ng/mL at all visits through

WK5D1 to WK25D1. Subjects who have no testosterone measurements

between WK5D1 and WK25D1 will be excluded from this analysis.

Frequency distributions will be provided for each treatment group. The

two-sided 95% confidence interval will also be provided.

## 4.3.2 Serum Concentrations of LH, FSH, DHT, and SHBG

Analysis Set: Full Analysis Set

Analysis

Variable(s): (1) Serum Concentrations of LH (mIU/mL)

(2) Serum Concentrations of FSH (mIU/mL)

(3) Serum Concentrations of DHT (ng/mL)

(4) Serum Concentrations of SHBG (nmol/L)

Visit: Baseline, WK1D2, WK1D4, WK2D1, WK3D1, WK5D1, WK9D1,

WK13D1, WK17D1, WK21D1, WK25D1, WK37D1, WK49D1, WK61D1,

# WK73D1, WK85D1, WK97D1

Analytical

Method(s):

The following analysis will be performed using the full analysis set. For the analysis variables (1) to (4), descriptive statistics of the observed values and the two-sided 95% confidence intervals of the mean will be provided for each visit by treatment group. The same analysis will be performed for the percent change from baseline. Case plots as well as the mean and standard deviation plots of changes over time will be provided for observed values for each treatment group.

#### 4.4 Statistical/Analytical Issues

## 4.4.1 Adjustments for Covariates

Not applicable in this study.

## 4.4.2 Handling of Dropouts or Missing Data

Missing test results and data determined to be non-evaluable according to the Handling Rules for Analysis Data will not be used for hypothesis testing and estimations.

Values less than or equal to the lower limit of quantification will be treated as the value of the lower limit of quantification for PSA, serum testosterone, high-sensitivity serum testosterone, LH, FSH, DHT, and SHBG, and all others will be treated as zero when calculating the descriptive statistics.

Values less than the lower limit of quantification will be treated as zero for the calculation of descriptive statistics except for geometric mean for plasma concentration of TAK-385. For the geometric mean, values less than the lower limit of quantification will be treated as missing.

## 4.4.3 Interim Analyses and Data Monitoring

No interim analysis is planned in this study.

### 4.4.4 Multicenter Studies

Although this study is a multicenter study, treatment-by-center interaction will not be explored since the number of subjects for each center is not sufficient for such exploration.

### 4.4.5 Multiple Comparison/Multiplicity

Not applicable in this study.

## 4.4.6 Use of an "Efficacy Subset" of Subjects

Not applicable in this study.

### 4.4.7 Active-Control Studies Intended to Show Equivalence or Non-Inferiority

Not applicable in this study.

## 4.4.8 Examination of Subgroups

Not applicable in this study.

#### 5 Safety Analysis (Part A)

In this study, safety will be evaluated as the primary endpoint.

#### **5.1 Treatment-Emergent Adverse Events**

Analysis will be performed on TEAEs that occurred in Part A.

## 5.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

Categories: Relationship to Study Drug [Related, Not Related]

Intensity [Grade 1, Grade 2, Grade 3, Grade 4, Grade 5]

Analytical

Method(s): The following summaries will be provided for each treatment group.

TEAEs will be graded using the National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

- (1) Overview of Treatment-Emergent Adverse Events
  - 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 2) Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
  - 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 6) Relationship of serious Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
  - Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 8) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

## Number of subjects

• Summaries for 2) and 6)

A subject with occurrences of TEAE in both categories (i.e., Related and

Not Related) will be counted once in the Related category.

• Summary for 3)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

• Summaries other than 2), 3), and 6)

A subject with multiple occurrences of TEAE will be counted only once.

## Number of events

For each summary, the total number of events will be calculated.

## 5.1.2 Displays of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

Categories: Intensity [Grade 1, Grade 2, Grade 3, Grade 4, Grade 5]

Time of Onset (day) [1 <= - <= 7, 8 <= - <= 14, 15 <= - <= 21,

 $22 \le - \le Max$ 

Analytical

Method(s): The following summaries will be provided using frequency distribution for each treatment group.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

TEAEs will be graded using the National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Drug-Related Treatment-Emergent Adverse Events by Preferred Term
- (6) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (7) Intensity of Drug-Related Treatment-Emergent Adverse Events by

- System Organ Class and Preferred Term
- (8) Treatment-Emergent Adverse Events with Intensity of Grade 3 or Higher by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (10) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (11) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (12) Special Interest Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

### Number of subjects

- Summary tables other than (6), (7), (8), and (11)
   A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.
- Summary tables for (6), (7), and (8)
   A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity.
   Percentages will be based on the number of subjects in the safety analysis set.
- Summary table for (11)

A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT.

When calculating percentages for each time interval, the number of subjects at risk (i.e., subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

### **5.1.3 Displays of Dose-Limiting Toxicities**

Analysis Set: DLT Analysis Set

Analysis

Variable(s): TEAE

Analytical

Method(s): The following summaries will be provided using frequency distribution for

each treatment group.

TEAEs considered as dose-limiting toxicities will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) Treatment-Emergent Adverse Events Considered as Dose-Limiting
Toxicities by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

## Number of subjects

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the DLT analysis set.

### **5.2 Pretreatment Events**

#### **5.2.1 Displays of Pretreatment Events**

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): PTE

Analytical

Method(s): The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Pretreatment Events by System Organ Class and Preferred Term
- (2) Serious Pretreatment Events by System Organ Class and Preferred Term Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

#### 5.3 Laboratory and Other Safety Data

## 5.3.1 Laboratory Test Results

## 5.3.1.1 Hematology, Biochemistry, and Lipid and Glycated Hemoglobin in Blood

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Hematology

Red Blood Cell White Blood Cell Hemoglobin

Hematocrit Platelets

Differential WBC (Neutrophils, Neutrophil Count, Basophils, Eosinophils,

Lymphocytes, Monocytes)

Biochemistry

Protein Total Albumin Glucose
Creatinine Blood Urea Uric Acid

Nitrogen

Bilirubin Total ALT (GPT) AST (GOT)

LDH GGT Alkaline Phosphatase

CK (CPK) Sodium Potassium

Chloride Calcium Corrected Calcium

Phosphorus PT-INR

Lipid and Glycated Hemoglobin in Blood

Triglycerides Total Cholesterol HDL Cholesterol

LDL Cholesterol TSH HbA1c

Categories: Intensity [Grade 0, Grade 1, Grade 2, Grade 3, Grade 4]

Visit: (1) and (2):

Hematology, Biochemistry: Baseline, D7, D14, D21, D28, SFU Lipid and Glycated Hemoglobin in Blood: Baseline, D28, SFU

Analytical

Method(s): For each variable, summaries (1) and (2) will be provided by treatment group.

For applicable variables, summaries (3), (4), and (5) will be provided by treatment group. Takeda Preferred SI Units will be used for all summaries.

(1) Summary of Laboratory Test Results and Change from Baseline by

Visit

Descriptive statistics for observed values and changes from baseline will be provided for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Number and Percentage of Subjects with Elevated Liver Enzyme

**Laboratory Parameters** 

Overall frequency distributions of elevated hepatic parameters will be provided. Further details are given in the Appendix.

- (4) Number and Percentage of Subjects with Laboratory Test Abnormalities by Grade
  - Frequency distributions for each laboratory test abnormality will be provided by grade. Evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data) obtained after baseline will be used. A subject with multiple occurrences of laboratory test abnormality will be counted once for the abnormality with the maximum intensity.
- (5) Maximum Grade Shift From Baseline of Laboratory Parameters The maximum post-baseline grade will be determined for each subject. Shift tables showing the number of subjects in each grade category at baseline and post-baseline visit will be provided using evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data).

### 5.3.1.2 Urinalysis

Analysis Set: Safety Analysis Set

Analysis

Variable(s): pH

Specific Gravity

Protein [-, +-, 1+, 2+, 3+, 4+, 5+]
Glucose [-, +-, 1+, 2+, 3+, 4+, 5+]
Occult blood [-, +-, 1+, 2+, 3+, 4+, 5+]
Ketones [-, +-, 1+, 2+, 3+, 4+, 5+]
Urobilinogen [-, +-, 1+, 2+, 3+, 4+, 5+]
Bilirubin [-, +-, 1+, 2+, 3+, 4+, 5+]

Categories: Intensity [Grade 0, Grade 1, Grade 2, Grade 3, Grade 4]

Visit: (1), (2), and (3): Baseline, D7, D14, D21, D28, SFU

Analytical

Method(s): For pH and specific gravity, summaries (1) and (2) will be provided by

treatment group.

For each variable other than pH and specific gravity, summary (3) will be provided by treatment group.

For protein, summaries (4) and (5) will also be provided by treatment group.

(1) Summary of Urine Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline will be provided for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

- (3) Number of Subjects in Categories of Urine Laboratory Test Results
  Shift tables showing the number of subjects in each category at baseline
  and each post-baseline visit will be provided.
- (4) Number and Percentage of Subjects with Urine Laboratory Test
  Abnormalities by Grade
  Frequency distributions for each urine laboratory test abnormality will
  be provided by grade. Evaluable data (i.e., non-missing and acceptable
  according to the Handling Rules for Analysis Data) obtained after
  baseline will be used. A subject with multiple occurrences of laboratory
  test abnormality will be counted once for the abnormality with the
- (5) Maximum Grade Shift From Baseline of Urine Laboratory Parameters The maximum post-baseline grade will be determined for each subject. Shift tables showing the number of subjects in each grade category at baseline and post-baseline visit will be provided using evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data).

### 5.3.2 Vital Signs, Physical Findings, and Other Observations Related to Safety

maximum intensity.

## 5.3.2.1 Vital Signs and Weight

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Body Temperature (C)

Systolic Blood Pressure (mmHg)
Diastolic Blood Pressure (mmHg)

Pulse (bpm)
Weight (kg)

Visit: (1) and (2): Baseline, D7, D14, D21, D28, SFU

Analytical

 $Method(s): \qquad \text{For each variable, summaries (1) and (2) will be provided by treatment group.}$ 

For applicable variables, summary (3) will be provided by treatment group.

(1) Summary of Vital Signs and Weight Parameters and Change from

Baseline by Visit

Descriptive statistics for observed values and changes from baseline will be provided for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Number and Percentage of Subjects with Markedly Abnormal Values of Vital Signs Parameters

Overall frequency distributions of MAV will be provided. If a vital sign parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

### 5.3.2.2 12-lead ECG

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Heart Rate (bpm)

RR Interval (msec)

PR Interval (msec)

QRS Interval (msec)

QT Interval (msec)

QTcF Interval (msec) observed value: [Min<= - <=449, 450<= - <=479,

 $480 \le -499,500 \le -400$ 

change from baseline:

 $[Min \le - \le 29, 30 \le - \le 59, 60 \le - \le Max]$ 

QTcB Interval (msec) observed value: [Min<= - <=449, 450<= - <=479,

 $480 \le -499,500 \le -400$ 

change from baseline:

 $[Min \le - \le 29, 30 \le - \le 59, 60 \le - \le Max]$ 

12-Lead ECG

Interpretation [Within Normal Limits, Abnormal but not

Clinically Significant, Abnormal and Clinically

Significant]

Visit: (1), (2), and (4): Baseline, D14, D28, SFU

Analytical

Method(s): For each variable other than 12-lead ECG interpretations, summaries (1) and

(2) will be provided by treatment group.

For applicable variables, summary (3) will be provided by treatment group.

For 12-lead ECG interpretation, summary (4) will be provided by treatment

group.

- (1) Summary of ECG Parameters and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline will be provided for each visit. Frequency distributions for the categorical variables will be provided for each visit.
- Case Plots
   Plots over time for each subject will be presented.
- (3) Number and Percentage of Subjects with Markedly Abnormal Values of ECG Parameters
  - Overall frequency distributions of MAV will be provided. If an ECG parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.
- (4) Summary of Shifts of ECG Parameters Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

## 5.4 Displays of Treatment-Emergent Adverse Events (Japanese)

Analysis Set: Safety Analysis Set

DLT Analysis Set

Analysis

Variable(s): TEAE

Analytical

Method(s): The following TEAEs will be summarized in the same way as in section 5.1.2 and section 5.1.3. All SOC and PT will be presented in Japanese.

- (1) Treatment-Emergent Adverse Events by Preferred Term
- (2) Drug-Related Treatment-Emergent Adverse Events by Preferred Term
- (3) Treatment-Emergent Adverse Events with Intensity of Grade 3 or Higher by System Organ Class and Preferred Term
- (4) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (5) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Treatment-Emergent Adverse Events Considered as Dose-Limiting Toxicities by System Organ Class and Preferred Term

#### 6 Safety Analysis (Part B)

In this study, safety will be evaluated as the primary endpoint.

#### **6.1 Treatment-Emergent Adverse Events**

Analysis will be performed on TEAEs that occurred in Part B.

## 6.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

Categories: Relationship to Study Drug [Re

[Related, Not Related]

Intensity [

[Grade 1, Grade 2, Grade 3, Grade 4, Grade 5]

Analytical

Method(s): The following summaries will be provided for each treatment group.

TEAEs will be graded using the National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

- (1) Overview of Treatment-Emergent Adverse Events
  - 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 2) Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
  - 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 6) Relationship of serious Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
  - Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 8) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

## Number of subjects

• Summaries for 2) and 6)

A subject with occurrences of TEAE in both categories (i.e., Related and

Not Related) will be counted once in the Related category.

• Summary for 3)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

• Summaries other than 2), 3), and 6)

A subject with multiple occurrences of TEAE will be counted only once.

## Number of events

For each summary, the total number of events will be calculated.

## 6.1.2 Displays of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

Categories: Intensity [Grade 1, Grade 2, Grade 3, Grade 4, Grade 5]

Time of Onset (day) [1 <= - <= 90, 91 <= - <= 180, 181 <= - <= 270,

271<= - <=360, 361<= - <=450, 451<= - <=540,

 $541 \le - \le 630, 631 \le - \le Max$ 

Analytical

Method(s): The following summaries will be provided using frequency distribution for each treatment group.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

TEAEs will be graded using the National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Drug-Related Treatment-Emergent Adverse Events by Preferred Term
- (6) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- (7) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (8) Treatment-Emergent Adverse Events with Intensity of Grade 3 or Higher by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (10) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (11) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (12) Special Interest Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

## Number of subjects

- Summary tables other than (6), (7), (8), and (11)
   A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.
- Summary tables for (6), (7), and (8)
   A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity.
   Percentages will be based on the number of subjects in the safety analysis set.
- Summary table for (11)

A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT.

When calculating percentages for each time interval, the number of subjects at risk (i.e., subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

#### **6.2 Pretreatment Events**

### **6.2.1 Displays of Pretreatment Events**

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): PTE

Analytical

Method(s): The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) Pretreatment Events by System Organ Class and Preferred Term

(2) Serious Pretreatment Events by System Organ Class and Preferred Term Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

#### 6.3 Laboratory and Other Safety Data

## 6.3.1 Laboratory Test Results

## 6.3.1.1 Hematology, Biochemistry, and Lipid and Glycated Hemoglobin in Blood

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Hematology

Red Blood Cell White Blood Cell Hemoglobin

Hematocrit Platelets

Differential WBC (Neutrophils, Neutrophil Count, Basophils, Eosinophils,

Lymphocytes, Monocytes)

Biochemistry

Protein Total Albumin Glucose
Creatinine Blood Urea Uric Acid

Nitrogen

Bilirubin Total ALT (GPT) AST (GOT)

LDH GGT Alkaline Phosphatase

CK (CPK) Sodium Potassium

Chloride Calcium Corrected Calcium

Phosphorus PT-INR

Lipid and Glycated Hemoglobin in Blood

Triglycerides Total Cholesterol HDL Cholesterol

LDL Cholesterol TSH HbA1c

Categories: Intensity [Grade 0, Grade 1, Grade 2, Grade 3, Grade 4]

Visit: (1) and (2):

Hematology: Baseline, WK5D1, WK9D1, WK13D1, WK25D1, WK37D1,

WK49D1, WK61D1, WK73D1, WK85D1, WK97D1, SFU

Biochemistry: Baseline, WK5D1, WK9D1, WK13D1, WK17D1, WK21D1,

WK25D1, WK29D1, WK33D1, WK37D1, WK41D1,

WK45D1, WK49D1, WK61D1, WK73D1, WK85D1,

WK97D1, SFU

Lipid and Glycated Hemoglobin in Blood:

Baseline, WK5D1, WK9D1, WK13D1, WK25D1, WK49D1,

WK61D1, WK73D1, WK85D1, WK97D1, SFU

Analytical

Method(s): For each variable, summaries (1) and (2) will be provided by treatment group.

For applicable variables, summaries (3), (4), and (5) will be provided by

treatment group. Takeda Preferred SI Units will be used for all summaries.

(1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline will be provided for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

- (3) Number and Percentage of Subjects with Elevated Liver Enzyme Laboratory Parameters
  - Overall frequency distributions of elevated hepatic parameters will be provided. Further details are given in Appendix.
- (4) Number and Percentage of Subjects with Laboratory Test Abnormalities by Grade
  - Frequency distributions for each laboratory test abnormality will be provided by grade. Evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data) obtained after baseline will be used. A subject with multiple occurrences of laboratory test abnormality will be counted once for the abnormality with the maximum intensity.
- (5) Maximum Grade Shift From Baseline of Laboratory Parameters The maximum post-baseline grade will be determined for each subject. Shift tables showing the number of subjects in each grade category at baseline and post-baseline visit will be provided using evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data).

## 6.3.1.2 Urinalysis

Analysis Set: Safety Analysis Set

Analysis

Variable(s): pH

Specific Gravity

Protein [-, +-, 1+, 2+, 3+, 4+, 5+]
Glucose [-, +-, 1+, 2+, 3+, 4+, 5+]
Occult blood [-, +-, 1+, 2+, 3+, 4+, 5+]
Ketones [-, +-, 1+, 2+, 3+, 4+, 5+]
Urobilinogen [-, +-, 1+, 2+, 3+, 4+, 5+]
Bilirubin [-, +-, 1+, 2+, 3+, 4+, 5+]

Categories: Intensity [Grade 0, Grade 1, Grade 2, Grade 3, Grade 4]

Visit: (1), (2), and (3):

Baseline, WK5D1, WK9D1, WK13D1, WK25D1, WK49D1, WK61D1, WK73D1, WK85D1, WK97D1, SFU

Analytical

Method(s): For pH and specific gravity, summaries (1) and (2) will be provided by treatment group.

For each variable other than pH and specific gravity, summary (3) will be provided by treatment group.

For protein, summaries (4) and (5) will also be provided by treatment group.

(1) Summary of Urine Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline will be provided for each visit.

- (2) Case PlotsPlots over time for each subject will be presented.
- (3) Number of Subjects in Categories of Urine Laboratory Test Results
  Shift tables showing the number of subjects in each category at baseline
  and each post-baseline visit will be provided.
- (4) Number and Percentage of Subjects with Urine Laboratory Test Abnormalities by Grade Frequency distributions for each urine laboratory test abnormality will be provided by grade. Evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data) obtained after baseline will be used. A subject with multiple occurrences of laboratory test abnormality will be counted once for the abnormality with the maximum intensity.
- (5) Maximum Grade Shift From Baseline of Urine Laboratory Parameters The maximum post-baseline grade will be determined for each subject. Shift tables showing the number of subjects in each grade category at baseline and post-baseline visit will be provided using evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data).

### 6.3.2 Vital Signs, Physical Findings, and Other Observations Related to Safety

### 6.3.2.1 Vital Signs and Weight

Analysis Set: Safety Analysis Set

**Analysis** 

Variable(s): Body Temperature (C)

Systolic Blood Pressure (mmHg)
Diastolic Blood Pressure (mmHg)

Pulse (bpm)
Weight (kg)

Visit: (1) and (2):

Baseline, WK2D1, WK3D1, WK5D1, WK9D1, WK13D1, WK25D1,

WK49D1, WK61D1, WK73D1, WK85D1, WK97D1, SFU

Analytical

Method(s): For each variable, summaries (1) and (2) will be provided by treatment group.

For applicable variables, summary (3) will be provided by treatment group.

(1) Summary of Vital Signs and Weight Parameters and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline will be provided for each visit.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Number and Percentage of Subjects with Markedly Abnormal Values of Vital Signs Parameters

Overall frequency distributions of MAV will be provided. If a vital sign parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

#### 6.3.2.2 12-lead ECG

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Heart Rate (bpm)

RR Interval (msec)
PR Interval (msec)
QRS Interval (msec)
QT Interval (msec)

QTcF Interval (msec) observed value: [Min<= - <=449, 450<= - <=479,

480<= - <=499, 500<= - <=Max]

change from baseline:

 $[Min \le - \le 29, 30 \le - \le 59, 60 \le - \le Max]$ 

QTcB Interval (msec) observed value: [Min<= - <=449, 450<= - <=479,

480<= - <=499, 500<= - <=Max]

change from baseline:

 $[Min \le - \le 29, 30 \le - \le 59, 60 \le - \le Max]$ 

12-Lead ECG

Interpretation [Within Normal Limits, Abnormal but not Clinically

Significant, Abnormal and Clinically Significant]

Visit: (1), (2), and (4):

Baseline, WK3D1, WK5D1, WK25D1, WK49D1, WK73D1, WK97D1, SFU

Analytical

Method(s): For each variable other than 12-lead ECG interpretations, summaries (1) and (2) will be provided by treatment group.

For applicable variables, summary (3) will be provided by treatment group. For 12-lead ECG interpretation, summary (4) will be provided by treatment group.

- (1) Summary of ECG Parameters and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline will be provided for each visit. Frequency distributions for the categorical variables will be provided for each visit.
- (2) Case PlotsPlots over time for each subject will be presented.
- (3) Number and Percentage of Subjects with Markedly Abnormal Values of ECG Parameters

Overall frequency distributions of MAV will be provided. If an ECG parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

(4) Summary of Shifts of ECG Parameters Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

### **6.3.2.3** Bone Mineral Density

Analysis Set: Safety Analysis Set

Analysis

Variable(s): (1) Bone Mineral Density ( $L_{2-4}$ )

(2) Bone Mineral Density (Femoral Neck)

(3) Bone Mineral Density (Total Hip)

Visit: Baseline, WK25D1, WK49D1, WK73D1, WK97D1

Analytical

Method(s): The following analysis will be performed using the safety analysis set.

For (1) to (3), the descriptive statistics of the observed values and the two-sided 95% confidence intervals of the mean will be provided for each visit by treatment group. The same analysis will be performed for the percent

change from baseline.

## 6.4 Displays of Treatment-Emergent Adverse Events (Japanese)

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

Analytical

Method(s): The following TEAEs will be summarized in the same way as in section

6.1.2. All SOC and PT will be presented in Japanese.

- (1) Treatment-Emergent Adverse Events by Preferred Term
- (2) Drug-Related Treatment-Emergent Adverse Events by Preferred Term
- (3) Treatment-Emergent Adverse Events with Intensity of Grade 3 or Higher by System Organ Class and Preferred Term
- (4) Treatment-Emergent Adverse Events Leading to Study Drug
  Discontinuation by System Organ Class and Preferred Term
- (5) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

## 7 Significance Level and Confidence Coefficient (Part A and Part B)

• Confidence coefficient: 95% (two-sided)

# **Amendment History**

| Version | Date | Author | Detailed Description of Amendments to Text |
|---|---|---|---|
| 1 | April 16, 2015 | | Not applicable |
| 2 | July 20, 2017 | | Refer to Appendix 1. |

Appendix 1. Amendments from the Previous Version

| Page | Existing Text | Revised Text | Rationale for Amendment |
|---|---|---|---|
| Cover | | | Updated in accordance with the |
| | | | current organization. |
| Cover | | | Updated in accordance with the |
| | | | current organization. |
| 4 | Glossary | Glossary | Added to clearly define the |
| | Descriptive statistics: number of subjects, mean, | Descriptive statistics: number of subjects, mean, | abbreviation. |
| | standard deviation, maximum, minimum, and quartiles | standard deviation (SD), maximum (max), minimum | |
| | | (min), and quartiles | |
| 4 | Glossary | Glossary | Added to clearly define the |
| | (New) | CV: coefficient of variation | abbreviation. |
| 4 | Glossary | Glossary | Added to clearly define the |
| | (New) | PK: pharmacokinetic | abbreviation. |
| 6 | Definition of Visit Window | Definition of Visit Window | Corrected to a more appropriate |
| | <part a=""> Pharmacokinetic Assessments</part> | <part a=""> Pharmacokinetic Assessments</part> | expression. |
| | Headers of the table: Visit, Scheduled Study Day | Headers of the table: Visit, Scheduled Study Time | |

| Page | Existing Text | Revised Text | Rationale for Amendment |
|---|---|---|---|
| | (days), Scheduled Study Time (hours), and Time | (hours), and Time Interval (Study Day (days), Study | |
| | Interval (Study Day (days), Study Time (hours)) | Time (hours)) | |
| 6 | Definition of Visit Window | Definition of Visit Window | Corrected to a more appropriate |
| | <part a=""> Pharmacokinetic Assessments</part> | <part a=""> Pharmacokinetic Assessments</part> | expression. |
| | | The visit windows in the whole table were revised. | |
| 11 | Definition of Visit Window | Definition of Visit Window | Corrected to a more appropriate |
| | <part b=""> Pharmacokinetic Assessments</part> | <part b=""> Pharmacokinetic Assessments</part> | expression. |
| | Headers of the table: Visit, Scheduled Study Day | Headers of the table: Visit, Scheduled Study Time | |
| | (days), Scheduled Study Time (hours), and Time | (hours), and Time Interval (Study Day (days), Study | |
| | Interval (Study Day (days), Study Time (hours)) | Time (hours)) | |
| 11 | Definition of Visit Window | Definition of Visit Window | Corrected to a more appropriate |
| | <part b=""> Pharmacokinetic Assessments</part> | <part b=""> Pharmacokinetic Assessments</part> | expression. |
| | | The visit windows in the whole table were revised. | |
| 20 | Others | Others | Corrected according to the latest |
| | PK parameters | The symbols and the definitions of PK parameter were | standard PK terminology |
| | | revised. | |
| 20 | Others | Others | Deleted unnecessary PK parameters |
| | AUC(0-inf)Area under the plasma/blood/serum | (deleted) | |
| | concentration-time curve from time 0 to infinity, | | |
| | calculated as AUC(0-inf)=AUC(0-tlqc)+lqc/λz, where | | |
| | tlqc is the time of last quantifiable concentration and | | |
| | lqc is the last quantifiable concentration. | | |

| Page | Existing Text | Revised Text | Rationale for Amendment |
|---|---|---|---|
| | AUMC(0-inf) Area under the first moment | | |
| | plasma/blood/serum concentration-time curve from | | |
| | time 0 to infinity, calculated as | | |
| | AUMC(0-inf)=AUMC(0-tlqc)+lqc $\times$ tlqc/ $\lambda$ z+lqc/ $\lambda$ z2, | | |
| | where tlqc is the time of last quantifiable concentration | | |
| | and lqc is the last quantifiable concentration. | | |
| 20 | Others | Others | Corrected to a more appropriate |
| | Cmax/DDose-adjusted Cmax. | $C_{max, ss}/D$ Dose-normalized $C_{max, ss}$ . | expression. |
| 20 | Others | Others | Deleted unnecessary PK parameters |
| | MRT Mean residence time, calculated as | (deleted) | |
| | MRT=AUMC(0-inf)/AUC(0-inf). | | |
| 20 | Others | Others | Corrected to a more appropriate |
| | Vss/FApparent volume of distribution at steady state | $V_z/F_{ss}$ Apparent volume of distribution during the | expression. |
| | after extravascular administration, calculated as Vss/F= | terminal disposition phase after extravascular | |
| | CL/F×MRT. | administration, calculated using $AUC_{\tau}$ | |
| 36 | 3.2.1 Plasma Concentrations | 3.2.1 Plasma Concentrations | Corrected to clarify which descriptive |
| | Descriptive statistics, geometric mean, and coefficient | Number of subjects, mean, SD, min, median, max, | statistics and linear plots will be |
| | of variation will be used to summarize plasma | geometric mean, and CV will be used to summarize | provided. |
| | concentrations at each visit. Plasma concentration-time | plasma concentrations at each visit for each treatment | |
| | profiles will be provided for each treatment group | group. | |
| | using individual or mean concentrations. | Linear plots of plasma concentration-time profiles will | |
| | | be provided for each treatment group using individual | |

| Page | Existing Text | Revised Text | Rationale for Amendment |
|---|---|---|---|
| | | and mean (SD) concentrations in separate plots. Mean | |
| | | (SD) plots will include the plasma concentration plot | |
| | | for all visits, separate plots for each of Day 1, Day 14, | |
| | | Day 28, and a plot for the plasma trough | |
| | | concentrations. | |
| 36 | (New) | Listing | Added to separate the listing for PK |
| | | Analysis Set: Full Analysis Set | parameters from the table of |
| | | Analysis Variable(s): | descriptive statistics. PK parameter |
| | | D1: AUC <sub><math>\tau</math></sub> , C <sub>max</sub> and t <sub>max</sub> | calculation methods were also moved |
| | | D14: $AUC_{last, SS}$ , $AUC_{\tau, SS}$ , $AUC_{\tau, SS}/D$ , $C_{max, SS}$ , $C_{max, SS}/D$ , | to this new section. |
| | | $C_{min, ss}, t_{max, ss}$ | |
| | | D28: $AUC_{last, SS}$ , $AUC_{\tau, SS}$ , $AUC_{\tau, SS}$ /D, $CL/F_{sS}$ , $C_{max, SS}$ , | |
| | | $C_{\text{max, ss}}/D$ , $t_{\text{max, ss}}$ , $t_{1/2z}$ , $V_z/F_{\text{ss}}$ , $\lambda_z$ , number of data points | |
| | | with first and last data points used in the terminal | |
| | | disposition phase regression analysis and adjusted R <sup>2</sup> | |
| | | (coefficient of determination) for the terminal | |
| | | disposition phase regression analysis | |
| | | Analytical Method(s): | |
| | | PK parameters will be calculated by using individual | |
| | | plasma concentrations with actual sampling times. | |
| | | Plasma concentrations from D1 to D2, D14 to D15 and | |
| | | D28 to D35 will be used for the calculation of PK | |

| Page | Existing Text | Revised Text | Rationale for Amendment |
|---|---|---|---|
| | | parameters on D1, D14 and D28 respectively. Plasma | |
| | | concentrations deviated from the visit window will be | |
| | | also used for the calculation. A standard | |
| | | non-compartmental analysis will be performed using | |
| | | the linear trapezoidal rule. If subject received | |
| | | prohibited concomitant medications, therapies or foods, | |
| | | then the plasma concentrations measured on and after | |
| | | this day will be used to estimate the PK parameters for | |
| | | the listing but the results will be treated as reference | |
| | | values. | |
| | | Individual PK parameters will be listed. The listings | |
| | | will include the treatment group, subject ID and | |
| | | evaluation day (D1, D14, and D28) in addition to the | |
| | | PK parameters. | |
| 37 | Descriptive Statistics | Descriptive Statistics | Added the dose-normalized PK |
| | D1: AUC(0-24), Cmax and Tmax | D1: AUC $_{\tau}$ , C <sub>max</sub> and t <sub>max</sub> | parameters ( $C_{max, ss}/D$ and $AUC_{\tau, ss}/D$ ) |
| | D14: AUC(0-tlqc), AUC(0-tau), AUC(0-tau)/D, Cmax, | D14: AUC <sub>last, ss</sub> , AUC <sub><math>\tau</math>, ss</sub> , AUC <sub><math>\tau</math>, ss</sub> /D, C <sub>max, ss</sub> , C <sub>max, ss</sub> | and corrected PK parameter symbols |
| | Cmax/D, Cmin, Tmax | ss/D, C <sub>min, ss</sub> , t <sub>max, ss</sub> | according to the latest standard PK |
| | D28: AUC(0-tlqc), AUC(0-tau), CL/F, Cmax, Tmax, | D28: AUC <sub>last, ss</sub> , AUC <sub><math>\tau</math>, ss</sub> , AUC <sub><math>\tau</math>, ss</sub> /D, CL/F <sub>ss</sub> , C <sub>max, ss</sub> , | terminology. |
| | T1/2, Vss/F | $C_{\text{max, ss}}/D$ , $t_{\text{max, ss}}$ , $t_{1/2z}$ , $V_z/F_{\text{ss}}$ , $\lambda_z$ | |
| 37 | Descriptive Statistics | Descriptive Statistics | Corrected to specify which |
| | Pharmacokinetic (PK) parameters will be calculated by | For the pharmacokinetic parameters, the number of | descriptive statistics will be provided. |

| Page | Existing Text | Revised Text | Rationale for Amendment |
|---|---|---|---|
| | using individual plasma concentrations with actual | subjects, mean, SD, min, median, max, geometric | The rules for data handling and the |
| | sampling times. Plasma concentrations from D1 to D2, | mean, and CV will be provided for each treatment | method for dose-proportionality |
| | D14 to D15 and D28 to D35 will be used for the | group. PK parameters which are treated as reference | assessment were changed to what |
| | calculation of PK parameters on D1, D14 and D28 | values will be excluded from the summary statistics. | was considered more appropriate. |
| | respectively. Plasma concentrations deviated from the | Graphical assessment of dose-proportionality on $C_{max}$ , | |
| | visit window will be also used for the calculation. A | $_{ss}$ and $AUC_{\tau, ss}$ will be conducted on D14 and D28 by | |
| | standard non-compartmental analysis will be | plotting individual dose-normalized exposure | |
| | performed. The listing of calculated PK parameters | parameters, i.e., $C_{max, ss}/D$ or $AUC_{\tau, ss}/D$ versus dose. | |
| | will be prepared for each subject. Descriptive statistics, | | |
| | geometric mean, and coefficient of variation will be | | |
| | used to summarize each pharmacokinetic parameter for | | |
| | each treatment group. Graphical assessment of | | |
| | dose-linearity on Cmax or AUC(0-tau) will be | | |
| | conducted on D14 and D28. | | |
| 39 | 3.4.2 Handling of Dropouts or Missing Data | 3.4.2 Handling of Dropouts or Missing Data | Added to define the rules for |
| | (New) | Values less than the lower limit of quantification will | handling values less than the lower |
| | | be treated as zero except for the calculation of | limit of quantification. |
| | | geometric mean for plasma concentration of TAK-385. | |
| | | For the geometric mean, values less than the lower | |
| | | limit of quantification will be treated as missing. | |
| 41 | 4.1.2 QOL Assessment | 4.1.2 QOL Assessment | Appendix containing details on the |
| | The following analysis will be performed using the full | The following analysis will be performed using the full | scoring procedures was added. |

| Page | Existing Text | Revised Text | Rationale for Amendment |
|---|---|---|---|
| | analysis set. | analysis set. The scoring procedures are described in | |
| | | detail in the Appendix. | |
| 41 | 4.2.1 Plasma Concentrations | 4.2.1 Plasma Concentrations | Corrected to a more appropriate |
| | Descriptive statistics, geometric mean, and coefficient | Descriptive statistics, geometric mean, and CV will be | expression. |
| | of variation will be used to summarize plasma | used to summarize plasma concentrations at each visit | |
| | concentrations at each visit. Plots of plasma | for each treatment group. Case plots as well as the | |
| | concentrations at each visit will be provided for each | mean and standard deviation plots of changes over time | |
| | treatment group using individual or mean | will be provided for plasma concentrations for each | |
| | concentrations. | treatment group. | |
| 42 | 4.3.1 Serum Testosterone Concentrations | 4.3.1 Serum Testosterone Concentrations | Added to align with other similar |
| | (2) High-sensitivity Serum Testosterone (ng/dL) | (2) High-sensitivity Serum Testosterone | expressions. |
| | | Concentrations (ng/dL) | |
| 42 | 4.3.1 Serum Testosterone Concentrations | 4.3.1 Serum Testosterone Concentrations | Added to clarify which analysis will |
| | Case plots as well as the mean and standard deviation | Case plots as well as the mean and standard deviation | include the reference line. |
| | plots of changes over time will be provided for | plots of changes over time will be provided for | |
| | observed values for each treatment group. A reference | observed values for each treatment group. For (1), a | |
| | line will be drawn where the serum testosterone | reference line will be drawn where the serum | |
| | concentration is 0.5 ng/mL. | testosterone concentration is 0.5 ng/mL. | |
| 44 | 4.4.2 Handling of Dropouts or Missing Data | 4.4.2 Handling of Dropouts or Missing Data | Added to define the rules for |
| | (New) | Values less than the lower limit of quantification will | handling values less than the lower |
| | | be treated as zero for the calculation of descriptive | limit of quantification. |
| | | statistics except for geometric mean for plasma | |

| Page | Existing Text | Revised Text | Rationale for Amendment |
|---|---|---|---|
| | | concentration of TAK-385. For the geometric mean, | |
| | | values less than the lower limit of quantification will be | |
| | | treated as missing. | |
| 65 | Appendix. Criteria for Markedly Abnormal Values and | Appendix 2. Criteria for Markedly Abnormal Values | Appendix number was updated since |
| | Elevated Liver Enzyme | and Elevated Liver Enzyme | Appendix 1 and 3 were added to the |
| | | | SAP. |
| 70 | (New) | Appendix 3. QOL Scoring Procedures | Added Appendix 3 to make clear of |
| | | | each of the QOL scoring procedures. |

## Appendix 2. Criteria for Markedly Abnormal Values and Elevated Liver Enzyme

### (1) Criteria for Markedly Abnormal Values

## 1) Vital Signs, and 12-lead ECG (except Upper MAV Criteria of QTcF Interval)

For each parameter, all evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data) obtained after baseline will be classified as a MAV or not. The criteria in the table below will be used. The lower limit of the normal range and the upper limit of the normal range are abbreviated as LLN and ULN.

Vital Signs

| | G . | Age | MAV Criteria | |
|---|---|---|---|---|
| Parameter | Gender | | Lower Criteria | Upper Criteria |
| Systolic Blood Pressure (mmHg) | - | - | <85 | >180 |
| Diastolic Blood Pressure (mmHg) | - | - | <50 | >110 |
| Pulse (bpm) | - | - | <50 | >120 |
| Body Temperature (°C) | - | - | <35.6 | >37.7 |

## 12-lead ECG

| | | r Age | MAV Criteria | |
|----------------------|--------|-------|----------------|----------------|
| Parameter | Gender | | Lower Criteria | Upper Criteria |
| Heart Rate (bpm) | - | - | <50 | >120 |
| QT Interval (msec) | - | - | <=50 | >=460 |
| QTcF Interval (msec) | - | - | <=50 | - |

## Classifying Subjects for the Overall Treatment Period

For each parameter and subject, classifications will be made according to the conditions i) to iii) provided below. The lower and the upper criteria will be considered separately.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that doesn't meet the MAV criteria will be considered as a subject without MAV.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV for that parameter.

## 2) 12-lead ECG (Upper MAV Criteria of QTcF Interval)

All evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data) obtained after baseline will be classified as a MAV or not. The criteria in the table below will be used. Note that the observed value and the change from baseline used for classification should be measurements taken on the same day.

| | a . | | MAV ( | Criteria |
|---|---|---|---|---|
| Parameter | Gender | Age | Lower Criteria | Upper Criteria |
| QTcF Interval (msec) | - | - | - | If either of the following conditions is met: - observed value >=500 - change from baseline >= 30 and observed value >=450 |

## Classifying Subjects for the Overall Treatment Period

For each subject, classifications will be made according to the conditions i) to iii) provided below.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that meets any of the following will be considered as a subject without MAV.
  - Observed value is less than 450 msec and not missing.
  - Change from baseline is less than 30 msec and not missing, and observed value is less than 500 msec and not missing.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV.

## (2) Criteria for Elevated Liver Enzyme

All evaluable data (i.e., non-missing and acceptable according to the Handling Rules for Analysis Data) obtained after baseline will be used to determine whether each criteria for elevated liver enzyme in the table below is met or not. If there is more than one parameter that need to be considered for a criteria, parameter measurements taken on the same day will be used. The following abbreviations are used: LLN for lower limit of the normal range, ULN for upper limit of the normal range, ALT for alanine aminotransferase, AST for aspartate aminotransferase, Tbili for total bilirubin, and ALP for alkaline phosphatase.

| | Criteria for Elevated Liver Enzyme | |
|---|---|---|
| Label | (a) Elevated | (b) Not Elevated |
| ALT > 3xULN | ALT is greater than 3 times the ULN | ALT is non-missing and less than or equal to 3 times the ULN |
| ALT > 5xULN | ALT is greater than 5 times the ULN | ALT is non-missing and less than or equal to 5 times the ULN ALT is non-missing and less than or equal to 8 times the ULN |
| ALT > 8xULN | ALT is greater than 8 times the ULN | |
| ALT > 3xULN with Tbili > 2xULN | ALT is greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | Either ALT is non-missing and less than or equal to 3 times the ULN, or the total bilirubin is non-missing and less than or equal to twice the ULN |
| AST > 3xULN | AST is greater than 3 times the ULN | AST is non-missing and less than or equal to 3 times the ULN |
| AST > 5xULN | AST is greater than 5 times the ULN | AST is non-missing and less than or equal to 5 times the ULN |
| AST > 8xULN | AST is greater than 8 times the ULN | AST is non-missing and less than or equal to 8 times the ULN |
| AST > 3xULN with Tbili > 2xULN | AST is greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | Either AST is non-missing and less than or equal to 3 times the ULN, or the total bilirubin is non-missing and less than or equal to twice the ULN |
| ALT or AST > 3xULN | Either ALT or AST is greater than 3 times the ULN | Both ALT and AST are non-missing and less than or equal to 3 times the ULN |
| ALT or AST > 5xULN | Either ALT or AST is greater than 5 times the ULN | Both ALT and AST are non-missing and less than or equal to 5 times the ULN |
| ALT or AST > 8xULN | Either ALT or AST is greater than 8 times | Both ALT and AST are non-missing and |

| T 1 1 | Criteria for Elevated Liver Enzyme | |
|---|---|---|
| Label | (a) Elevated | (b) Not Elevated |
| | the ULN | less than or equal to 8 times the ULN |
| ALT or AST > 3xULN | Either ALT or AST is greater than 3 times | If any of the following conditions is met: - Both ALT and AST are non-missing and |
| | the ULN and the total bilirubin is greater | less than or equal to 3 times the ULN. |
| with Tbili > 2xULN | than twice the ULN | - Total bilirubin is non-missing and less |
| | | than or equal to twice the ULN. |
| | | Either ALT is non-missing and less than |
| | Both ALT and AST are greater than 3 | or equal to 3 times the ULN, or AST is |
| ALT and AST > 3xULN | times the ULN | non-missing and less than or equal to 3 |
| | | times the ULN |
| | | Either ALT is non-missing and less than |
| ALT and AST > 5xULN | Both ALT and AST are greater than 5 | or equal to 5 times the ULN, or AST is |
| ALI and ASI > SAULIN | times the ULN | non-missing and less than or equal to 5 |
| | | times the ULN |
| | | Either ALT is non-missing and less than |
| ALT and AST > 8xULN | Both ALT and AST are greater than 8 | or equal to 8 times the ULN, or AST is |
| | times the ULN | non-missing and less than or equal to 8 |
| | | times the ULN |
| | | If any of the following conditions is met: |
| | | - ALT is non-missing and less than or |
| ALT and AST > 3xULN | Both ALT and AST are greater than 3 | equal to 3 times the ULN |
| with Tbili > 2xULN | times the ULN and the total bilirubin is | - AST is non-missing and less than or |
| | greater than twice the ULN | equal to 3 times the ULN |
| | | - Total bilirubin is non-missing and less<br>than or equal to twice the ULN |
| | ALP is greater than 3 times the ULN | ALP is non-missing and less than or equal |
| ALP > 3xULN | | to 3 times the ULN |
| | | Either ALP is non-missing and less than or |
| | | equal to 3 times the ULN, or ALT is |
| ALP > 3xULN | Both ALP and ALT are greater than 3 | non-missing and less than or equal to 3 |
| with ALT > 3xULN | time the ULN | times the ULN |
| ALP > 3xULN | Both ALP and AST are greater than 3 | Either ALP is non-missing and less than or |

| | Criteria for Elevated Liver Enzyme | |
|---|---|---|
| Label | (a) Elevated | (b) Not Elevated |
| with AST > 3xULN | times the ULN | equal to 3 times the ULN, or AST is |
| | | non-missing and less than or equal to 3 |
| | | times the ULN |

## **Appendix 3. QOL Scoring Procedures**

### (1) AMS

AMS subscale scores and total scores will be calculated as follows. If one or more of the scores required for the calculation of a subscale are missing, then that particular subscale and the total score will be treated as missing.

- Psychological subscale: sum of severity points from questions 6, 7, 8, 11, 13
- Somatic subscale: sum of severity points from questions 1, 2, 3, 4, 5, 9, 10
- Sexual subscale: sum of severity points from questions 12, 14, 15, 16, 17
- Total score: sum of severity points from all questions from 1 to 17

Reference: Moore C, Huebler D, Zimmermann T, Heinemann LA, Saad F, Thai DM. The Aging Males' Symptoms scale (AMS) as outcome measure for treatment of androgen deficiency. Eur Urol 2004;46(1):80-7

### (2) EORTC QLQ-C30

The Global health status/QoL score and each Functional scales score (physical, role, emotional, cognitive, social) will be calculated as follows. The "range" used in the calculations is the difference between the maximum possible values of the score and the minimum possible value. If more than half of the scores are missing, then the Global health status/QoL score or the Functional scales score will be treated as missing. If at least half of the scores are available, then the scores that are available will be used for the calculation.

- Global health status/QoL score: {[(average of item 29 & 30)-1]/range}\*100
- Physical functioning: {1-[(average of item 1 to 5)-1]/range}\*100
- Role functioning: {1-[(average of item 6 & 7)-1]/range}\*100
- Emotional functioning: {1-[(average of item 21 to 24)-1]/range}\*100
- Cognitive functioning: {1-[(average of item 20 & 25)-1]/range}\*100
- Social functioning: {1-[(average of item 26 & 27)-1]/range}\*100

Reference: Fayers PM, Aaronson NK, Bjordal K, Groenvold M, Curran D, Bottomley A, on behalf of the EORTC Quality of Life Group. *The EORTC QLQ-C30 Scoring Manual (3<sup>rd</sup> edition)*. Published by: European Organisation for Research and Treatment of Cancer, Brussels 2001.

## (3) EPIC

Each of the HRQOL Domain Summary Scores (urinary, bowel, sexual, hormonal) will be calculated according to the following steps.

1) Convert score using the conversion table below.

Conversion Table

| Converted Converted | | |
|---|---|---|
| Question No. | Answer | Converted<br>Score |
| 1, 2, 3, 8, 9, 14, 20, 21, 22, 23, 26, 27, 28, 29, 32 | 1 | 0 |
| | 2 | 25 |
| | 3 | 50 |
| | 4 | 75 |
| | 5 | 100 |
| 4 | 1 | 0 |
| | 2 | 33 |
| | 3 | 67 |
| | 4 | 100 |
| 5 | 0 | 100 |
| | 1 | 67 |
| | 2 | 33 |
| | 3 | 0 |
| 6A, 6B, 6C, 6D, 6E, 6F, 15A, 15B, 15C, 15D, | 0 | 100 |
| 15E, 15F, 24A, 24B, 24C, 31A, 31B, 31C, 31D, | 1 | 100 |
| 31E, 31F | 2 | 75 |
| | 3 | 50 |
| | 4 | 25 |
| | 5 | 0 |
| 7, 10, 11, 12, 16, 25 | 1 | 100 |
| | 2 | 75 |
| | 3 | 50 |
| | 4 | 25 |
| | 5 | 0 |
| 13 | 1 | 100 |
| | 2 | 50 |
| | 3 | 0 |
| 17A, 17B, 17C, 19 | 0 | 0 |
| | 1 | 0 |
| | 2 | 25 |
| | 3 | 50 |
| | 4 | 75 |
| | 5 | 100 |
| 18 | 0 | 0 |
| | 1 | 0 |
| | 2 | 33 |
| | 3 | 67 |
| | 4 | 100 |
| 30 | 1 | 0 |
| | 2 | 50 |
| | 3 | 100 |
| | 4 | 50 |
| | 5 | 0 |

- 2) Each of the HRQOL Domain Summary Scores (urinary, bowel, sexual, hormonal) will be calculated as follows. If 20% or more of the answers are missing then the summary score will not be calculated.
  - Urinary summary score: average of converted scores of question no. 1 to 7
  - Bowel summary score: average of converted scores of question no. 8 to 16
  - Sexual summary score: average of converted scores of question no. 17 to 25
  - Hormonal summary score: average of converted scores of question no. 26 to 31

Reference: Takegami M, Suzukamo Y, iHope International. EPIC. 2002.